CLINICAL TRIAL: NCT04090957
Title: A Randomized Double-blind Placebo Controlled Phase 3 Trial to Evaluate the Efficacy and Safety of Estetrol for the Treatment of Moderate to Severe Vasomotor Symptoms in Postmenopausal Women (E4Comfort Study II)
Brief Title: Estetrol for the Treatment of Moderate to Severe Vasomotor Symptoms in Postmenopausal Women (E4Comfort II)
Acronym: E4Comfort II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Estetra (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIT-Do001-C302
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Results first posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Vasomotor Symptoms; Menopausal Symptoms
Keywords: Estetrol; Hot Flushes; Vasomotor symptoms
MeSH Terms: conditions — Hot Flashes | interventions — Estetrol

STUDY DESIGN:
Intervention Model Description: For the Efficacy study part, there are 3 blinded arms (randomized) and for the Safety study part, there is 1 open-label (non-randomized) arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: There are 3 blinded arms in the Efficacy part and 1 open-labeled arm in the Safety part.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Estetrol 15 mg - Efficacy Study Part (Experimental): Estetrol (E4) 15 mg, administered orally once daily for up to 53 weeks.
  Interventions: Drug: Estetrol oral tablet
- Estetrol 20 mg - Efficacy Study Part (Experimental): Estetrol (E4) 20 mg, administered orally once daily for up to 53 weeks.
  Interventions: Drug: Estetrol oral tablet
- Placebo - Efficacy Study Part (Placebo Comparator): Placebo, administered orally once daily for up to 53 weeks.
  Interventions: Drug: Placebo oral tablet
- Estetrol 20 mg - Safety Study Part (Experimental): Estetrol (E4) 20 mg, administered orally once daily for up to 53 weeks.
  Interventions: Drug: Estetrol oral tablet

INTERVENTIONS:
Drug: Estetrol oral tablet — Estetrol oral tablet, administered orally once daily.
  Other Names: E4 oral tablet
  Arms: Estetrol 15 mg - Efficacy Study Part; Estetrol 20 mg - Efficacy Study Part; Estetrol 20 mg - Safety Study Part
Drug: Placebo oral tablet — Placebo oral tablet, administered orally once daily.
  Arms: Placebo - Efficacy Study Part

SUMMARY:
A two-part study designed to evaluate the effect of Estetrol (E4) 15 mg, 20 mg, or placebo on the severity and frequency of vasomotor symptoms (VMS) in the Efficacy Study Part and the safety of E4 20 mg in the Safety Study Part.

DETAILED DESCRIPTION:
This is a two-part study:

Arm 1, 2, and 3: randomized, double blind

- Efficacy Study Part: designed to evaluate the frequency and severity of vasomotor symptoms [VMS] in both hysterectomized and non hysterectomized postmenopausal participants after treatment with two doses of E4 (15 mg or 20 mg) or placebo for 12 consecutive weeks. Thereafter, treatment proceeded for a total duration of up to 53 weeks, to continue the evaluation of secondary efficacy (effect on hemostasis, lipid and glucose metabolism, bone turnover, health-related quality of life [HRQoL] and treatment satisfaction [TS]), safety and the effect on the endometrium. For endometrial protection, all non-hysterectomized subjects received 200 mg progesterone (P4) once daily for 14 consecutive days, after completion of the E4/placebo treatment.

Arm 4: open label

- Safety Study Part: designed to evaluate the general safety, secondary efficacy (lipid and glucose metabolism, HRQoL and TS) after treatment with E4 20 mg for up to 53 weeks in hysterectomized and non hysterectomized postmenopausal participants. For endometrial protection, all non-hysterectomized subjects received 200 mg progesterone (P4) once daily for 14 consecutive days, after completion of the E4 treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent form and any required privacy authorization prior to the initiation of any trial procedure, after the nature of the trial has been explained according to local regulatory requirements;
2. Females ≥ 40 up to ≤ 65 years of age at randomization/treatment allocation;
3. For hysterectomized subjects: documented hysterectomy must have occurred at least 6 weeks prior to the start of screening. Hysterectomy can be total or subtotal (i.e., cervix was not removed).
4. For non-hysterectomized subjects: uterus with bi-layer endometrial thickness ≤ 4 mm on transvaginal ultrasound (TVUS)
5. For non-hysterectomized subjects: endometrial biopsy taken during screening that reveals no abnormal result, i.e., presence of hyperplasia (simple or complex, with or without atypia), presence of carcinoma, and presence of disordered proliferative endometrium findings. The screening biopsy should have sufficient endometrial tissue for diagnosis. Biopsies without tissue or with insufficient tissue may be repeated once;
6. Seeking treatment for relief of VMS associated with menopause;

   1. For the Efficacy Study part: at least 7 moderate to severe bothersome VMS per day or at least 50 moderate to severe bothersome VMS per week in the last 7 consecutive days during the Screening period;
   2. For the Safety Study part: at least 1 moderate to severe VMS per week;
7. Body mass index ≥ 18.0 kg/m² up to ≤ 38.0 kg/m²;
8. A mammogram that shows no sign of significant disease performed during screening or within 9 months prior to the start of screening;
9. Post-menopausal status defined as any of the following:

   1. For non-hysterectomized subjects:

      * At least 12 months of spontaneous amenorrhea with serum follicle stimulating hormone (FSH) >40 milli-International unit (mIU)/mL (value obtained after washout of estrogen/progestin containing drugs, see exclusion criteria 18 and 20);
      * or at least 6 months of spontaneous amenorrhea with serum FSH >40 mIU /mL and E2 <20 pg/mL (value obtained after washout of estrogen/progestin containing drugs, see exclusion criteria 18 and 20);
      * or at least 6 weeks postsurgical bilateral oophorectomy;
   2. For hysterectomized subjects:

      * serum FSH >40 mIU/mL and E2 <20 pg/mL (values obtained after washout of estrogen/progestin containing drug, see exclusion criteria 18 and 20);
      * or at least 6 weeks post-surgical bilateral oophorectomy;
10. Good physical and mental health, in the judgement of the Investigator as based on medical history, physical and gynecological examination, and clinical assessments performed prior to Visit 1;
11. Able to understand and comply with the protocol requirements, instructions, and protocol-stated restrictions;
12. Able and willing to complete trial daily diaries and questionnaires.

Exclusion Criteria:

1. History of malignancy, with the exception of basal cell or squamous cell carcinoma of the skin if diagnosed more than 1 year prior to the Screening visit;
2. Any clinically significant findings found by the Investigator at the breast examination and/or on mammography suspicious of breast malignancy that would require additional clinical testing to rule out breast cancer (however, simple cysts confirmed by ultrasound are allowed);
3. Papanicolaou (PAP) test with atypical squamous cells undetermined significance (ASC-US) or higher (low-grade squamous intraepithelial lesion [LSIL], atypical squamous cells- cannot exclude high-grade squamous intraepithelial lesion [HSIL] [ASC-H], HSIL dysplastic or malignant cells) in sub-totally hysterectomized and non-hysterectomized subjects. Note: ASC-US is allowed if a reflex human papilloma virus (HPV) testing is performed and is negative for high risk oncogene HPV subtypes 16 and 18;
4. For non-hysterectomized subjects:

   1. History or presence of uterine cancer, endometrial hyperplasia, or disordered proliferative endometrium;
   2. Presence of endometrial polyp;
   3. Undiagnosed vaginal bleeding or undiagnosed abnormal uterine bleeding;
   4. Endometrial ablation;
   5. Any uterine/endometrial abnormality that in the judgment of the investigator contraindicates the use of estrogen and/or progestin therapy. This includes presence or history of adenomyosis or significant myoma;
5. Systolic blood pressure (BP) higher than 130 mmHg, diastolic BP higher than 80 mmHg during screening;
6. History of venous or arterial thromboembolic disease (e.g., superficial or deep vein thrombosis, pulmonary embolism, stroke, myocardial infarction, angina pectoris, etc.), or first-degree family history of venous thromboembolism (VTE);
7. History of known acquired of congenital coagulopathy or abnormal coagulation factors, including known thrombophilia's;
8. Laboratory values of fasting glucose above 125 mg/dL and/or glycated hemoglobin above 7%;
9. Dyslipoproteinaemia (LDL >190 mg/dL and/or triglycerides >300 mg/dL);
10. Subjects smoking >15 cigarettes per day;
11. Presence or history of gallbladder disease, unless cholecystectomy has been performed;
12. Systemic lupus erythematosus;
13. Any malabsorption disorders including gastric bypass surgery;
14. History of acute liver disease in the preceding 12 months before the start of screening or presence or history of chronic or severe liver disease [alanine transaminase (ALT) or aspartate transaminase (AST) >2 x upper limit of normal (ULN), bilirubin >1.5 ULN], or liver tumors;
15. Chronic or current acute renal impairment (estimated glomerular filtration rate <60 ml/min);
16. Porphyria;
17. Diagnosis or treatment of major psychiatric disorder (e.g., schizophrenia, bipolar disorder, etc.) in the judgement of the Investigator;
18. Use of estrogen/progestin containing drug(s) up to:

    1. 1 week before screening start for vaginal non-systemic hormonal products (rings, creams, gels);
    2. 4 weeks before screening start for vaginal or transdermal estrogen or estrogen/progestin products;
    3. 8 weeks before screening start for oral estrogen and/or progestin products and/or selective estrogen receptor modulator therapy;
    4. 8 weeks before screening start for intrauterine progestin therapy;
    5. 3 months before screening start for progestin implants or estrogen alone injectable drug therapy;
    6. 6 months before screening start for estrogen pellet therapy or progestin injectable drug therapy;
19. Use of androgen/dehydroepiandrosterone (DHEA) containing drugs:

    1. 8 weeks before screening start for oral, topical, vaginal or transdermal androgen;
    2. 6 months before screening start for implantable or injectable androgen therapy;
20. Use of phytoestrogens or black cohosh for treatment of VMS up to 2 weeks before the start of screening;
21. For the women participating in the Efficacy Study part: use of prescription or over-the-counter products used for the treatment of VMS, e.g., anti-depressants: paroxetine, escitalopram, methyldopa, opioid and clonidine up to 4 weeks before the start of screening, and venlafaxine and desvenlafaxine up to 3 months before the start of screening , and not willing to stop these during their participation in the trial;
22. Not willing to stop any hormonal products as described in exclusion criteria 18, 19 and 20 during their participation in the trial;
23. Inadequately treated hyperthyroidism with abnormal thyroid stimulating hormone (TSH) and free T4 at screening. Subjects with low or high TSH are allowed if free T4 at screening is within normal range;
24. History or presence of allergy/intolerance to the investigational product or drugs of this class or any component of it, or history of drug or other allergy that, in the opinion of the Investigator contraindicates subject participation;
25. For non-hysterectomized subjects: history or presence of allergy to peanuts;
26. History of alcohol or substance abuse (including marijuana, even if legally allowed) or dependence in the previous 12 months before the start of screening as determined by the Investigator, based on reported observations;
27. Sponsor or contract research organization (CRO) employees or employees under the direct supervision of the Investigator and/or involved directly in the trial;
28. Subjects with known or suspected history of a clinically significant systemic disease, unstable medical disorders, life-threatening disease or current malignancies that would pose a risk to the subject in the opinion of the Investigator;
29. Participation in another investigational drug clinical trial within 1 month (30 days) or having received an investigational drug within the last month (30 days) before the start of screening;
30. Is judged by the Investigator to be unsuitable for any reason.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1015 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Estetra, Study Director — Estetra
Locations (90):
- United States (85):
  - Estetra Study Site, Birmingham, Alabama
  - Estetra Study Site, Dothan, Alabama
  - Estetra Study Site, Phoenix, Arizona
  - Estetra Study Site, Tempe, Arizona
  - Estetra Study Site, Tucson, Arizona
  - Estetra Study Site, Little Rock, Arkansas
  - Estetra Study Site, Bellflower, California
  - Estetra Study Site, Canoga Park, California
  - Estetra Study Site, Chula Vista, California
  - Estetra Study Site, Huntington Beach, California
  - Estetra Study Site, La Mesa, California
  - Estetra Study Site, Lincoln, California
  - Estetra Study Site, Los Angeles, California
  - Estetra Study Site, Pomona, California
  - Estetra Study Site, Sacramento, California
  - Estetra Study Site, San Diego, California
  - Estetra Study Site, Santa Ana, California
  - Estetra Study Site, Thousand Oaks, California
  - Estetra Study Site, West Covina, California
  - Estetra Study Site, Colorado Springs, Colorado
  - Estetra Study Site, Denver, Colorado
  - Estetra Study Site, Crystal River, Florida
  - Estetra Study Site, Jacksonville, Florida
  - Estetra Study Site, Miami, Florida
  - Estetra Study Site, Miami Lakes, Florida
  - Estetra Study Site, New Port Richey, Florida
  - Estetra Study Site, Ocoee, Florida
  - Estetra Study Site, Orlando, Florida
  - Estetra Study Site, Sarasota, Florida
  - Estetra Study Site, West Palm Beach, Florida
  - Estetra Study Site, Atlanta, Georgia
  - Estetra Study Site, Morrow, Georgia
  - Estetra Study Site, Sandy Springs, Georgia
  - Estetra Study Site, Savannah, Georgia
  - Estetra Study Site, Idaho Falls, Idaho
  - Estetra Study Site, Meridian, Idaho
  - Estetra Study Site, Evansville, Indiana
  - Estetra Study Site, Marrero, Louisiana
  - Estetra Study Site, Saginaw, Michigan
  - Estetra Study Site, Rochester, Minnesota
  - Estetra Study Site, St Louis, Missouri
  - Estetra Study Site, Lincoln, Nebraska
  - Estetra Study Site, Norfolk, Nebraska
  - Estetra Study Site, Las Vegas, Nevada
  - Estetra Study Site, Albuquerque, New Mexico
  - Estetra Study Site, New York, New York
  - Estetra Study Site, Charlotte, North Carolina
  - Estetra Study Site, Columbus, North Carolina
  - Estetra Study Site, Fayetteville, North Carolina
  - Estetra Study Site, Hickory, North Carolina
  - Estetra Study Site, New Bern, North Carolina
  - Estetra Study Site, Raleigh, North Carolina
  - Estetra Study Site, Rocky Mount, North Carolina
  - Estetra Study Site, Cincinnati, Ohio
  - Estetra Study Site, Cleveland, Ohio
  - Estetra Study Site, Columbus, Ohio
  - Estetra Study Site, Fairfield, Ohio
  - Estetra Study Site, Erie, Pennsylvania
  - Estetra Study Site, Philadelphia, Pennsylvania
  - Estetra Study Site, Bluffton, South Carolina
  - Estetra Study Site, Columbia, South Carolina
  - Estetra Study Site, Mt. Pleasant, South Carolina
  - Estetra Study Site, Myrtle Beach, South Carolina
  - Estetra Study Site, North Charleston, South Carolina
  - Estetra Study Site, Chattanooga, Tennessee
  - Estetra Study Site, Jefferson City, Tennessee
  - Estetra Study Site, Knoxville, Tennessee
  - Estetra Study Site, Memphis, Tennessee
  - Estetra Study Site, Dallas, Texas
  - Estetra Study Site, Fort Worth, Texas
  - Estetra Study Site, Georgetown, Texas
  - Estetra Study Site, Houston, Texas
  - Estetra Study Site, McAllen, Texas
  - Estetra Study Site, Pearland, Texas
  - Estetra Study Site, Plano, Texas
  - Estetra Study Site, San Antonio, Texas
  - Estetra Study Site, Draper, Utah
  - Estetra Study Site, Pleasant Grove, Utah
  - Estetra Study Site, West Jordan, Utah
  - Estetra Study Site, Charlottesville, Virginia
  - Estetra Study Site, Norfolk, Virginia
  - Estetra Study Site, Virginia Beach, Virginia
  - Estetra Study Site, Bellevue, Washington
  - Estetra Study Site, Seattle, Washington
  - Estetra Study Site, Morgantown, West Virginia
- Canada (5):
  - Estetra Study Site, Red Deer, Alberta
  - Estetra Study Site, Montreal, Quebec
  - Estetra Study Site, Brampton
  - Estetra Study Site, Québec
  - Estetra Study Site, Waterloo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Panay N, Simoncini T, Taziaux M, Bouchard C, Black A, Kapoor E, Utian W, Foidart JM, Lobo RA. Estetrol for the treatment of moderate to severe vasomotor symptoms in postmenopausal women: The design of the E4COMFORT I and II trials. Maturitas. 2026 Jan;204:108781. doi: 10.1016/j.maturitas.2025.108781. Epub 2025 Nov 17. PMID 41289787

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment process for the overall study involved hysterectomized and non hysterectomized postmenopausal women ≥40 up to ≤65 years of age seeking treatment for the relief of vasomotor symptoms (VMS) associated with menopause; N=3974 were screened by study inclusion and exclusion criteria.
  * Efficacy Study Part: >=7 moderate to severe VMS/day or >=50 moderate to severe VMS/week in the last 7 consecutive days during the screening period.
  * Safety Study Part: >=1 moderate to severe VMS/week.
Groups:
- Estetrol 15 mg - Randomized Set - Efficacy Study Part: Estetrol monohydrate 15 mg (E4 15 mg), equivalent to estetrol 14.2 mg. The study drug was to be taken once a day for up to 53 weeks.
- Estetrol 20 mg - Randomized Set - Efficacy Study Part; Estetrol 20 mg - Included Set - Safety Study Part: Estetrol monohydrate 20 mg (E4 20 mg), equivalent to estetrol 18.9 mg. The study drug was to be taken once a day for up to 53 weeks.
- Placebo - Randomized Set - Efficacy Study Part: Placebo was administered orally once daily for up to 53 weeks.
Period: Overall Study
Arm/Group | Estetrol 15 mg - Randomized Set - Efficacy Study Part | Estetrol 20 mg - Randomized Set - Efficacy Study Part | Placebo - Randomized Set - Efficacy Study Part | Estetrol 20 mg - Included Set - Safety Study Part
Started | 194 | 194 | 196 | 431
Completed | 96 | 85 | 108 | 149
Not Completed | 98 | 109 | 88 | 282
Not completed — Lost to Follow-up | 22 | 25 | 25 | 36
Not completed — Withdrawal of Consent for Another Reason | 15 | 17 | 21 | 39
Not completed — Adverse Event | 19 | 25 | 8 | 104
Not completed — Other | 10 | 6 | 5 | 12
Not completed — Serious Adverse Event | 7 | 11 | 1 | 32
Not completed — Endometrial Biopsy Showing Proliferative Disorder | 7 | 9 | 1 | 26
Not completed — Lack of Efficacy | 1 | 1 | 9 | 0
Not completed — Protocol Violation | 3 | 5 | 2 | 1
Not completed — Withdrawal of Consent Due to Lack of Efficacy | 2 | 2 | 6 | 3
Not completed — COVID-19 | 2 | 2 | 3 | 7
Not completed — Non-Compliance with Trial Protocol: Other | 2 | 2 | 1 | 4
Not completed — Physician Decision | 2 | 1 | 1 | 5
Not completed — Sponsor Decision | 1 | 1 | 1 | 3
Not completed — Endometrial Findings - Physician Decision | 1 | 1 | 0 | 5
Not completed — Non-Compliance to Trial Protocol: Study Drug Intake Compliance | 1 | 0 | 1 | 4
Not completed — Non-Compliance to Trial Protocol: VMS Count Compliance | 0 | 0 | 1 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — No Treatment Administered | 2 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Arms 1-3 Safety Analysis Set (SAF): consisted of all randomized subjects who received at least one dose of randomized study medication. The SAF was used for all safety analyses and background characteristics and all analyses on this set were based on the treatment received.
  Arm 4 Safety Analysis Set (SAF): included all subjects who received at least one dose of study medication. The SAF was used for all analyses of safety and background characteristics.
Groups:
- Estetrol 15 mg - Efficacy Study Part: Estetrol (E4) 15 mg oral tablet, administered once daily for up to 53 weeks
- Estetrol 20 mg - Efficacy Study Part; Estetrol 20 mg - Safety Study Part: Estetrol (E4) 20 mg oral tablet, administered once daily for up to 53 weeks
- Placebo - Efficacy Study Part: Placebo was administered orally once daily for up to 53 weeks.
- Total: Total of all reporting groups
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part | Estetrol 20 mg - Safety Study Part | Total
Number analyzed (Participants) | 192 | 193 | 194 | 430 | 1009
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (5.14) | 54.5 (4.83) | 54.7 (4.68) | 54.4 (4.88) | 54.7 (4.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 192 | 193 | 194 | 430 | 1009
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 74 | 59 | 66 | 83 | 282
  Not Hispanic or Latino | 118 | 134 | 128 | 347 | 727
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 3 | 0 | 4
  Asian | 1 | 3 | 1 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 54 | 55 | 50 | 95 | 254
  White | 136 | 133 | 139 | 325 | 733
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 1 | 4 | 7
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.83 (4.59) | 27.93 (4.40) | 28.75 (4.61) | 28.33 (4.54) | 28.43 (4.545)
Education Level [Count of Participants; unit: Participants]
  Less than Upper Secondary School | 5 | 6 | 11 | 6 | 28
  Completed Upper Secondary School | 57 | 68 | 49 | 126 | 300
  Completed Vocational School | 32 | 23 | 25 | 42 | 122
  Completed College | 71 | 73 | 81 | 204 | 429
  Completed Graduate School | 22 | 19 | 26 | 46 | 113
  Unknown | 5 | 4 | 2 | 6 | 17
Smoking status at screening [Count of Participants; unit: Participants] — Population: Results shown for subjects with available data.
  Participants
    YES, Hysterectomized: number analyzed (Participants) | 99 | 100 | 99 | 201 | 499
    YES, Hysterectomized | 9 | 8 | 9 | 24 | 50
    YES, Non-Hysterectomized: number analyzed (Participants) | 93 | 93 | 95 | 229 | 510
    YES, Non-Hysterectomized | 6 | 14 | 9 | 27 | 56
    NO, Hysterectomized: number analyzed (Participants) | 99 | 100 | 99 | 201 | 499
    NO, Hysterectomized | 90 | 92 | 90 | 177 | 449
    NO, Non-Hysterectomized: number analyzed (Participants) | 93 | 93 | 95 | 229 | 510
    NO, Non-Hysterectomized | 87 | 79 | 86 | 202 | 454
Cigarettes smoked per day [Count of Participants; unit: Participants] — Population: Results shown for subjects with available data.
  Participants
    ≤5, Hysterectomized: number analyzed (Participants) | 99 | 100 | 99 | 201 | 499
    ≤5, Hysterectomized | 7 | 4 | 5 | 11 | 27
    >5 - 15, Hysterectomized: number analyzed (Participants) | 99 | 100 | 99 | 201 | 499
    >5 - 15, Hysterectomized | 2 | 4 | 4 | 13 | 23
    >15, Hysterectomized: number analyzed (Participants) | 99 | 100 | 99 | 201 | 499
    >15, Hysterectomized | 0 | 0 | 0 | 0 | 0
    ≤5, Non-Hysterectomized: number analyzed (Participants) | 93 | 93 | 95 | 229 | 510
    ≤5, Non-Hysterectomized | 4 | 9 | 5 | 13 | 31
    >5 - 15, Non-Hysterectomized: number analyzed (Participants) | 93 | 93 | 95 | 229 | 510
    >5 - 15, Non-Hysterectomized | 1 | 5 | 4 | 14 | 24
    >15, Non-Hysterectomized: number analyzed (Participants) | 93 | 93 | 95 | 229 | 510
    >15, Non-Hysterectomized | 1 | 0 | 0 | 0 | 1
Hysterectomy [Count of Participants; unit: Participants]
  YES | 99 | 100 | 99 | 201 | 499
  NO | 93 | 93 | 95 | 229 | 510
Hysterectomy Type [Count of Participants; unit: Participants]
  Total | 79 | 67 | 69 | 138 | 353
  Subtotal | 20 | 33 | 30 | 63 | 146
Bilateral Oophorectomy [Count of Participants; unit: Participants]
  YES, Hysterectomized | 42 | 31 | 26 | 65 | 164
  NO, Hysterectomized | 57 | 69 | 73 | 136 | 335
  YES, Non-Hysterectomized | 0 | 0 | 0 | 0 | 0
  NO, Non-Hysterectomized | 93 | 93 | 95 | 229 | 510

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Weekly Frequency of Moderate to Severe Vasomotor Symptoms (VMS) From Baseline to Week 4 and Week 12 -- (Efficacy Study Part)
Description: Weekly frequency of moderate to severe VMS at Baseline = total number (sum) of all recorded moderate to severe VMS experienced during the last 7 consecutive days prior randomization (Week 0).
  Weekly frequency of moderate to severe VMS at Week X = total number (sum) of all recorded moderate to severe VMS experienced during the week X.
Time Frame: Week 0 (Baseline), Week 4, Week 12.
Population: Intention-to-treat (ITT) Set: included all subjects who received at least one dose of randomized study medication.
  The ITT set was the primary analysis set for the efficacy analyses and all analyses on this set were based on the randomized treatment.
Measure: Mean (95% Confidence Interval); unit: number of moderate to severe VMS
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
number of moderate to severe VMS
  Week 4: number analyzed (Participants) | 172 | 179 | 179
  Week 4 | -39.77 [-45.75 to -33.79] | -40.11 [-45.51 to -34.71] | -31.82 [-36.96 to -26.67]
  Week 12: number analyzed (Participants) | 156 | 153 | 150
  Week 12 | -55.84 [-63.58 to -48.09] | -59.47 [-66.98 to -51.95] | -43.27 [-48.82 to -37.71]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 4; E4 15 mg vs Placebo; Test type: Superiority; p = 0.0436, Mixed Model for Repeated Measures; Least square mean difference = -8.42, 95% CI 2-sided [-16.64 to -0.20]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 4; E4 20 mg vs Placebo; Test type: Superiority; p = 0.0117, Mixed Model for Repeated Measures; Least square mean difference = -10.21, 95% CI 2-sided [-18.44 to -1.98]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 12; E4 15 mg vs Placebo; Test type: Superiority; p = 0.0029, Mixed Model for Repeated Measures; Least square mean difference = -12.20, 95% CI 2-sided [-20.69 to -3.71]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 12; E4 20 mg vs Placebo; Test type: Superiority; p = 0.0001, Mixed Model for Repeated Measures; Least square mean difference = -15.49, 95% CI 2-sided [-24.04 to -6.94]

2. Primary Outcome: Mean Change in Severity of Moderate to Severe Vasomotor Symptoms (VMS) From Baseline to Week 4 and Week 12 -- (Efficacy Study Part)
Description: Mean severity score of VMS at Baseline: arithmetic mean of daily severity score values of moderate and severe VMS during the last 7 days prior randomization (Week 0). Mean severity score of VMS at Week 4 or 12: arithmetic mean of daily severity score values of moderate and severe VMS during Week 4 or 12.
  Daily severity score of VMS at Baseline = [(2 x number of moderate VMS) + (3 x number of severe VMS)]/(total number of moderate + severe VMS)], if at least one moderate to severe VMS was recorded during the day. If documented absence of moderate to severe VMS during the day, daily severity was set to zero.
  Daily severity score of VMS Post-Baseline = [(1 x number of mild VMS) + (2 x number of moderate VMS) + (3 x number of severe VMS)]/(total number of mild + moderate + severe VMS)], if at least one mild to severe VMS was recorded during the day. If documented absence of VMS during the day, daily severity was set to zero.
  Severity score: mild=1, moderate=2, severe=3.
Time Frame: Week 0 (Baseline), Week 4, Week 12.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
score
  Week 4: number analyzed (Participants) | 172 | 179 | 179
  Week 4 | -0.58 [-0.66 to -0.49] | -0.63 [-0.71 to -0.54] | -0.52 [-0.60 to -0.44]
  Week 12: number analyzed (Participants) | 156 | 153 | 150
  Week 12 | -0.77 [-0.87 to -0.66] | -1.01 [-1.13 to -0.88] | -0.73 [-0.85 to -0.62]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 4; E4 15 mg vs Placebo; Test type: Superiority; p = 0.7786, Mixed Model for Repeated Measures; Least square mean difference = -0.04, 95% CI 2-sided [-0.20 to 0.12]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 4; E4 20 mg vs Placebo; Test type: Superiority; p = 0.0310, Mixed Model for Repeated Measures; Least square mean difference = -0.17, 95% CI 2-sided [-0.33 to -0.01]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 12; E4 15 mg vs Placebo; Test type: Superiority; p = 0.7941, Mixed Model for Repeated Measures; Least square mean difference = -0.04, 95% CI 2-sided [-0.21 to 0.12]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 12; E4 20 mg vs Placebo; Test type: Superiority; p < .0001, Mixed Model for Repeated Measures; Least square mean difference = -0.35, 95% CI 2-sided [-0.51 to -0.18]

3. Secondary Outcome: Mean Change From Baseline to Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 in the Weekly Frequency of Moderate to Severe Vasomotor Symptoms (VMS) -- (Efficacy Study Part)
Description: Mean change from Baseline to Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 in the weekly frequency of moderate to severe vasomotor symptoms (VMS) (Efficacy study part).
  Weekly frequency of moderate to severe VMS at Baseline = total number (sum) of all recorded moderate to severe VMS experienced during the last 7 consecutive days prior randomization (Week 0).
  Weekly frequency of moderate to severe VMS at Week X = total number (sum) of all recorded moderate to severe VMS experienced during the week X.
Time Frame: Week 0 (Baseline), Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: number of moderate to severe VMS
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
number of moderate to severe VMS
  Week 1: number analyzed (Participants) | 172 | 183 | 181
  Week 1 | -16.20 [-21.36 to -11.03] | -18.00 [-22.38 to -13.62] | -15.62 [-20.42 to -10.81]
  Week 2: number analyzed (Participants) | 171 | 183 | 182
  Week 2 | -26.97 [-32.31 to -21.63] | -27.51 [-32.73 to -22.30] | -25.26 [-30.55 to -19.97]
  Week 3: number analyzed (Participants) | 172 | 180 | 181
  Week 3 | -34.60 [-40.05 to -29.14] | -34.99 [-40.58 to -29.40] | -29.47 [-34.81 to -24.13]
  Week 4: number analyzed (Participants) | 172 | 179 | 179
  Week 4 | -39.77 [-45.75 to -33.79] | -40.11 [-45.51 to -34.71] | -31.82 [-36.96 to -26.67]
  Week 5: number analyzed (Participants) | 169 | 174 | 173
  Week 5 | -42.98 [-49.18 to -36.78] | -46.68 [-52.82 to -40.55] | -35.14 [-40.80 to -29.49]
  Week 6: number analyzed (Participants) | 168 | 168 | 168
  Week 6 | -46.75 [-53.11 to -40.39] | -50.14 [-57.09 to -43.20] | -37.53 [-43.49 to -31.58]
  Week 7: number analyzed (Participants) | 165 | 165 | 167
  Week 7 | -48.78 [-55.58 to -41.99] | -51.95 [-59.05 to -44.85] | -38.39 [-44.23 to -32.55]
  Week 8: number analyzed (Participants) | 165 | 162 | 167
  Week 8 | -50.39 [-57.32 to -43.47] | -54.08 [-61.17 to -46.98] | -39.53 [-45.64 to -33.43]
  Week 9: number analyzed (Participants) | 160 | 162 | 160
  Week 9 | -53.94 [-61.77 to -46.11] | -55.79 [-62.57 to -49.01] | -40.87 [-46.41 to -35.33]
  Week 10: number analyzed (Participants) | 157 | 158 | 154
  Week 10 | -56.57 [-64.37 to -48.76] | -57.24 [-64.55 to -49.92] | -42.41 [-47.77 to -37.04]
  Week 11: number analyzed (Participants) | 157 | 155 | 154
  Week 11 | -55.81 [-63.63 to -48.00] | -58.12 [-65.63 to -50.60] | -41.81 [-47.28 to -36.34]
  Week 12: number analyzed (Participants) | 156 | 153 | 150
  Week 12 | -55.84 [-63.58 to -48.09] | -59.47 [-66.98 to -51.95] | -43.27 [-48.82 to -37.71]

4. Secondary Outcome: Mean Change in Severity of Moderate and Severe Vasomotor Symptoms (VMS) From Baseline to Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 -- (Efficacy Study Part)
Description: Mean severity score of VMS at Baseline: arithmetic mean of daily severity score values of moderate and severe VMS during the last 7 days prior randomization (Week 0). Mean severity score of VMS at Week X (post-baseline): arithmetic mean of daily severity score values of moderate and severe VMS during Week X.
  Daily severity score of VMS at Baseline = [(2 x number of moderate VMS) + (3 x number of severe VMS)]/(total number of moderate + severe VMS)], if at least one moderate to severe VMS was recorded during the day. If documented absence of moderate to severe VMS during the day, daily severity was set to zero.
  Daily severity score of VMS Post-Baseline = [(1 x number of mild VMS) + (2 x number of moderate VMS) + (3 x number of severe VMS)]/(total number of mild + moderate + severe VMS)], if at least one mild to severe VMS was recorded during the day. If documented absence of VMS during the day, daily severity was set to zero.
  Severity score: mild=1, moderate=2, severe=3.
Time Frame: Week 0 (Baseline), Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
score
  Week 1: number analyzed (Participants) | 172 | 183 | 181
  Week 1 | -0.30 [-0.35 to -0.24] | -0.31 [-0.36 to -0.25] | -0.33 [-0.37 to -0.28]
  Week 2: number analyzed (Participants) | 171 | 183 | 182
  Week 2 | -0.40 [-0.47 to -0.33] | -0.40 [-0.47 to -0.33] | -0.43 [-0.50 to -0.36]
  Week 3: number analyzed (Participants) | 172 | 180 | 181
  Week 3 | -0.51 [-0.59 to -0.42] | -0.57 [-0.65 to -0.48] | -0.49 [-0.57 to -0.41]
  Week 4: number analyzed (Participants) | 172 | 179 | 179
  Week 4 | -0.58 [-0.66 to -0.49] | -0.63 [-0.71 to -0.54] | -0.52 [-0.60 to -0.44]
  Week 5: number analyzed (Participants) | 169 | 174 | 173
  Week 5 | -0.63 [-0.73 to -0.53] | -0.72 [-0.82 to -0.62] | -0.54 [-0.63 to -0.45]
  Week 6: number analyzed (Participants) | 168 | 168 | 168
  Week 6 | -0.65 [-0.75 to -0.55] | -0.78 [-0.89 to -0.68] | -0.63 [-0.72 to -0.53]
  Week 7: number analyzed (Participants) | 165 | 165 | 167
  Week 7 | -0.65 [-0.75 to -0.56] | -0.88 [-0.99 to -0.76] | -0.64 [-0.73 to -0.54]
  Week 8: number analyzed (Participants) | 165 | 162 | 167
  Week 8 | -0.68 [-0.78 to -0.58] | -0.89 [-1.01 to -0.78] | -0.69 [-0.79 to -0.59]
  Week 9: number analyzed (Participants) | 160 | 162 | 160
  Week 9 | -0.76 [-0.87 to -0.66] | -0.91 [-1.02 to -0.79] | -0.66 [-0.76 to -0.56]
  Week 10: number analyzed (Participants) | 157 | 158 | 154
  Week 10 | -0.78 [-0.88 to -0.68] | -0.96 [-1.09 to -0.84] | -0.69 [-0.80 to -0.58]
  Week 11: number analyzed (Participants) | 157 | 155 | 154
  Week 11 | -0.79 [-0.89 to -0.68] | -0.96 [-1.08 to -0.83] | -0.68 [-0.80 to -0.56]
  Week 12: number analyzed (Participants) | 156 | 153 | 150
  Week 12 | -0.77 [-0.87 to -0.66] | -1.01 [-1.13 to -0.88] | -0.73 [-0.85 to -0.62]

5. Secondary Outcome: Mean Change From Baseline to Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 in the Weekly Frequency of Mild to Severe Vasomotor Symptoms (VMS) -- (Efficacy Study Part)
Description: Weekly frequency of mild to severe VMS at Baseline = total number (sum) of all recorded mild to severe VMS experienced during the last 7 consecutive days prior randomization (Week 0).
  Weekly frequency of mild to severe VMS at Week X = total number (sum) of all recorded mild to severe VMS experienced during the week X.
Time Frame: Week 0 (Baseline), Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: number of mild, moderate to severe VMS
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
number of mild, moderate to severe VMS
  Week 1: number analyzed (Participants) | 172 | 183 | 181
  Week 1 | -17.25 [-22.95 to -11.56] | -19.35 [-23.96 to -14.75] | -16.92 [-22.29 to -11.56]
  Week 2: number analyzed (Participants) | 171 | 183 | 182
  Week 2 | -28.20 [-34.15 to -22.24] | -28.88 [-34.47 to -23.28] | -28.47 [-34.37 to -22.57]
  Week 3: number analyzed (Participants) | 172 | 180 | 181
  Week 3 | -34.81 [-41.23 to -28.39] | -36.98 [-43.17 to -30.80] | -32.50 [-38.87 to -26.12]
  Week 4: number analyzed (Participants) | 172 | 179 | 179
  Week 4 | -40.49 [-47.34 to -33.63] | -43.12 [-49.18 to -37.07] | -35.18 [-41.62 to -28.73]
  Week 5: number analyzed (Participants) | 169 | 174 | 173
  Week 5 | -44.36 [-51.58 to -37.15] | -49.73 [-56.47 to -42.99] | -40.20 [-47.23 to -33.16]
  Week 6: number analyzed (Participants) | 168 | 168 | 168
  Week 6 | -48.24 [-55.84 to -40.64] | -53.27 [-60.86 to -45.68] | -42.95 [-50.27 to -35.64]
  Week 7: number analyzed (Participants) | 165 | 165 | 167
  Week 7 | -50.12 [-58.01 to -42.23] | -55.22 [-62.94 to -47.50] | -43.18 [-50.35 to -36.01]
  Week 8: number analyzed (Participants) | 165 | 162 | 167
  Week 8 | -52.04 [-60.25 to -43.83] | -57.42 [-65.21 to -49.63] | -44.32 [-51.75 to -36.90]
  Week 9: number analyzed (Participants) | 160 | 162 | 160
  Week 9 | -57.09 [-66.65 to -47.53] | -59.72 [-67.30 to -52.14] | -46.57 [-53.71 to -39.42]
  Week 10: number analyzed (Participants) | 157 | 158 | 154
  Week 10 | -59.91 [-69.64 to -50.17] | -61.75 [-69.83 to -53.67] | -48.50 [-55.72 to -41.28]
  Week 11: number analyzed (Participants) | 157 | 155 | 154
  Week 11 | -59.40 [-69.24 to 49.57] | -62.86 [-71.13 to -54.60] | -48.48 [-55.77 to -41.19]
  Week 12: number analyzed (Participants) | 156 | 153 | 150
  Week 12 | -59.78 [-69.41 to -50.14] | -64.76 [-73.24 to -56.29] | -49.03 [-56.44 to -41.62]

6. Secondary Outcome: Percentage of Subjects With ≥50% and ≥75% Reduction From Baseline in the Weekly Frequency of Moderate to Severe Vasomotor Symptoms (VMS) at Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 -- (Efficacy Study Part)
Description: Weekly frequency of moderate to severe VMS at Baseline = total number (sum) of all recorded moderate to severe VMS experienced during the last 7 consecutive days prior randomization (Week 0).
  Weekly frequency of moderate to severe VMS at Week X = Total number (sum) of all recorded moderate to severe VMS experienced during the week X
  Percentages of participants are based on the number of subjects with a non-missing percent change from Baseline result in each treatment arm by visit in the ITT Set.
Time Frame: Week 0 (Baseline), Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
percentage of participants
  Week 1: ≥50% reduction from baseline: number analyzed (Participants) | 171 | 183 | 181
  Week 1: ≥50% reduction from baseline | 17.0 | 20.8 | 17.1
  Week 1: ≥75% reduction from baseline: number analyzed (Participants) | 171 | 183 | 181
  Week 1: ≥75% reduction from baseline | 5.8 | 4.4 | 5.0
  Week 2: ≥50% reduction from baseline: number analyzed (Participants) | 170 | 183 | 182
  Week 2: ≥50% reduction from baseline | 31.2 | 31.7 | 29.1
  Week 2: ≥75% reduction from baseline: number analyzed (Participants) | 170 | 183 | 182
  Week 2: ≥75% reduction from baseline | 14.1 | 13.1 | 14.3
  Week 3: ≥50% reduction from baseline: number analyzed (Participants) | 171 | 180 | 181
  Week 3: ≥50% reduction from baseline | 42.7 | 44.4 | 37.6
  Week 3: ≥75% reduction from baseline: number analyzed (Participants) | 171 | 180 | 181
  Week 3: ≥75% reduction from baseline | 18.1 | 23.9 | 19.3
  Week 4: ≥50% reduction from baseline: number analyzed (Participants) | 171 | 179 | 179
  Week 4: ≥50% reduction from baseline | 51.5 | 53.6 | 44.1
  Week 4: ≥75% reduction from baseline: number analyzed (Participants) | 171 | 179 | 179
  Week 4: ≥75% reduction from baseline | 24.6 | 29.1 | 17.9
  Week 5: ≥50% reduction from baseline: number analyzed (Participants) | 168 | 174 | 173
  Week 5: ≥50% reduction from baseline | 57.7 | 64.4 | 46.8
  Week 5: ≥75% reduction from baseline: number analyzed (Participants) | 168 | 174 | 173
  Week 5: ≥75% reduction from baseline | 29.2 | 39.1 | 22.5
  Week 6: ≥50% reduction from baseline: number analyzed (Participants) | 167 | 168 | 168
  Week 6: ≥50% reduction from baseline | 61.7 | 70.2 | 51.8
  Week 6: ≥75% reduction from baseline: number analyzed (Participants) | 167 | 168 | 168
  Week 6: ≥75% reduction from baseline | 31.1 | 46.4 | 32.1
  Week 7: ≥50% reduction from baseline: number analyzed (Participants) | 164 | 165 | 167
  Week 7: ≥50% reduction from baseline | 62.2 | 70.9 | 55.1
  Week 7: ≥75% reduction from baseline: number analyzed (Participants) | 164 | 165 | 167
  Week 7: ≥75% reduction from baseline | 35.4 | 49.7 | 31.7
  Week 8: ≥50% reduction from baseline: number analyzed (Participants) | 164 | 162 | 167
  Week 8: ≥50% reduction from baseline | 64.0 | 70.4 | 55.7
  Week 8: ≥75% reduction from baseline: number analyzed (Participants) | 164 | 162 | 167
  Week 8: ≥75% reduction from baseline | 36.0 | 52.5 | 31.7
  Week 9: ≥50% reduction from baseline: number analyzed (Participants) | 159 | 162 | 160
  Week 9: ≥50% reduction from baseline | 75.5 | 74.1 | 58.8
  Week 9: ≥75% reduction from baseline: number analyzed (Participants) | 159 | 162 | 160
  Week 9: ≥75% reduction from baseline | 40.3 | 51.9 | 35.0
  Week 10: ≥50% reduction from baseline: number analyzed (Participants) | 156 | 158 | 154
  Week 10: ≥50% reduction from baseline | 76.9 | 78.5 | 64.3
  Week 10: ≥75% reduction from baseline: number analyzed (Participants) | 156 | 158 | 154
  Week 10: ≥75% reduction from baseline | 46.8 | 53.2 | 39.0
  Week 11: ≥50% reduction from baseline: number analyzed (Participants) | 156 | 155 | 154
  Week 11: ≥50% reduction from baseline | 78.8 | 80.0 | 62.3
  Week 11: ≥75% reduction from baseline: number analyzed (Participants) | 156 | 155 | 154
  Week 11: ≥75% reduction from baseline | 48.7 | 52.3 | 33.8
  Week 12: ≥50% reduction from baseline: number analyzed (Participants) | 155 | 153 | 150
  Week 12: ≥50% reduction from baseline | 81.3 | 81.7 | 61.3
  Week 12: ≥75% reduction from baseline: number analyzed (Participants) | 155 | 153 | 150
  Week 12: ≥75% reduction from baseline | 49.0 | 56.9 | 37.3
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 1, ≥50% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.9666, Chi-squared; Risk Difference (RD) = -0.2, 95% CI 2-sided [-8.0 to 7.7]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 1, ≥50% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.3759, Chi-squared; Risk Difference (RD) = 3.6, 95% CI 2-sided [-4.4 to 11.7]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 1, ≥75% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.7164, Chi-squared; Risk Difference (RD) = 0.9, 95% CI 2-sided [-3.9 to 5.6]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 1, ≥75% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.7859, Chi-squared; Risk Difference (RD) = -0.6, 95% CI 2-sided [-4.9 to 3.7]
Statistical Analysis 5: Comparison: Estetrol 15 mg - Efficacy Study Part vs Estetrol 20 mg - Efficacy Study Part; 5_Week 2, ≥50% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.6744, Chi-squared; Risk Difference (RD) = 2.1, 95% CI 2-sided [-7.5 to 11.6]
Statistical Analysis 6: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 6_Week 2, ≥50% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.5931, Chi-squared; Risk Difference (RD) = 2.6, 95% CI 2-sided [-6.9 to 12.0]
Statistical Analysis 7: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 7_Week 2, ≥75% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.9640, Chi-squared; Risk Difference (RD) = -0.2, 95% CI 2-sided [-7.5 to 7.1]
Statistical Analysis 8: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 8_Week 2, ≥75% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.7449, Chi-squared; Risk Difference (RD) = -1.2, 95% CI 2-sided [-8.2 to 5.9]
Statistical Analysis 9: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 9_Week 3, ≥50% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.3271, Chi-squared; Risk Difference (RD) = 5.1, 95% CI 2-sided [-5.1 to 15.4]
Statistical Analysis 10: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 10_Week 3, ≥50% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.1842, Chi-squared; Risk Difference (RD) = 6.9, 95% CI 2-sided [-3.2 to 17.0]
Statistical Analysis 11: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 11_Week 3, ≥75% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.7716, Chi-squared; Risk Difference (RD) = -1.2, 95% CI 2-sided [-9.4 to 6.9]
Statistical Analysis 12: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 12_Week 3, ≥75% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.2934, Chi-squared; Risk Difference (RD) = 4.6, 95% CI 2-sided [-3.9 to 13.0]
Statistical Analysis 13: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 13_Week 4, ≥50% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.1701, Chi-squared; Risk Difference (RD) = 7.3, 95% CI 2-sided [-3.1 to 17.8]
Statistical Analysis 14: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 14_Week 4, ≥50% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.0723, Chi-squared; Risk Difference (RD) = 9.5, 95% CI 2-sided [-0.8 to 19.8]
Statistical Analysis 15: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 15_Week 4, ≥75% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.1258, Chi-squared; Risk Difference (RD) = 6.7, 95% CI 2-sided [-1.9 to 15.2]
Statistical Analysis 16: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 16_Week 4, ≥75% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.0126, Chi-squared; Risk Difference (RD) = 11.2, 95% CI 2-sided [2.5 to 19.9]
Statistical Analysis 17: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 17_Week 5, ≥50% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.0436, Chi-squared; Risk Difference (RD) = 10.9, 95% CI 2-sided [0.4 to 21.5]
Statistical Analysis 18: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 18_Week 5, ≥50% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.0010, Chi-squared; Risk Difference (RD) = 17.5, 95% CI 2-sided [7.3 to 27.8]
Statistical Analysis 19: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 19_Week 5, ≥75% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.1623, Chi-squared; Risk Difference (RD) = 6.6, 95% CI 2-sided [-2.7 to 15.9]
Statistical Analysis 20: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 20_Week 5, ≥75% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.0009, Chi-squared; Risk Difference (RD) = 16.5, 95% CI 2-sided [7.0 to 26.1]
Statistical Analysis 21: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 21_Week 6, ≥50% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.0677, Chi-squared; Risk Difference (RD) = 9.9, 95% CI 2-sided [-0.7 to 20.4]
Statistical Analysis 22: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 22_Week 6, ≥50% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.0005, Chi-squared; Risk Difference (RD) = 18.5, 95% CI 2-sided [8.2 to 28.7]
Statistical Analysis 23: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 23_Week 6, ≥75% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.8432, Chi-squared; Risk Difference (RD) = -1.0, 95% CI 2-sided [-11.0 to 9.0]
Statistical Analysis 24: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 24_Week 6, ≥75% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.0073, Chi-squared; Risk Difference (RD) = 14.3, 95% CI 2-sided [4.0 to 24.6]
Statistical Analysis 25: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 25_Week 7, ≥50% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.1894, Chi-squared; Risk Difference (RD) = 7.1, 95% CI 2-sided [-3.5 to 17.7]
Statistical Analysis 26: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 26_Week 7, ≥50% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.0028, Chi-squared; Risk Difference (RD) = 15.8, 95% CI 2-sided [5.6 to 26.1]
Statistical Analysis 27: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 27_Week 7, ≥75% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.4844, Chi-squared; Risk Difference (RD) = 3.6, 95% CI 2-sided [-6.5 to 13.8]
Statistical Analysis 28: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 28_Week 7, ≥75% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.0009, Chi-squared; Risk Difference (RD) = 18.0, 95% CI 2-sided [7.6 to 28.4]
Statistical Analysis 29: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 29_Week 8, ≥50% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.1220, Chi-squared; Risk Difference (RD) = 8.3, 95% CI 2-sided [-2.2 to 18.9]
Statistical Analysis 30: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 30_Week 8, ≥50% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.0058, Chi-squared; Risk Difference (RD) = 14.7, 95% CI 2-sided [4.4 to 25.0]
Statistical Analysis 31: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 31_Week 8, ≥75% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.4151, Chi-squared; Risk Difference (RD) = 4.2, 95% CI 2-sided [-5.9 to 14.4]
Statistical Analysis 32: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 32_Week 8, ≥75% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.0001, Chi-squared; Risk Difference (RD) = 20.7, 95% CI 2-sided [10.3 to 31.2]
Statistical Analysis 33: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 33_Week 9, ≥50% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.0015, Chi-squared; Risk Difference (RD) = 16.7, 95% CI 2-sided [6.6 to 26.9]
Statistical Analysis 34: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 34_Week 9, ≥50% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.0036, Chi-squared; Risk Difference (RD) = 15.3, 95% CI 2-sided [5.1 to 25.5]
Statistical Analysis 35: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 35_Week 9, ≥75% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.3330, Chi-squared; Risk Difference (RD) = 5.3, 95% CI 2-sided [-5.4 to 15.9]
Statistical Analysis 36: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 36_Week 9, ≥75% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.0023, Chi-squared; Risk Difference (RD) = 16.9, 95% CI 2-sided [6.2 to 27.5]
Statistical Analysis 37: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 37_Week 10, ≥50% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.0146, Chi-squared; Risk Difference (RD) = 12.6, 95% CI 2-sided [2.6 to 22.7]
Statistical Analysis 38: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 38_Week 10, ≥50% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.0055, Chi-squared; Risk Difference (RD) = 14.2, 95% CI 2-sided [4.3 to 24.1]
Statistical Analysis 39: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 39_Week 10, ≥75% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.1635, Chi-squared; Risk Difference (RD) = 7.8, 95% CI 2-sided [-3.1 to 18.8]
Statistical Analysis 40: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 40_Week 10, ≥75% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.0119, Chi-squared; Risk Difference (RD) = 14.2, 95% CI 2-sided [3.3 to 25.2]
Statistical Analysis 41: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 41_Week 11, ≥50% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.0014, Chi-squared; Risk Difference (RD) = 16.5, 95% CI 2-sided [6.5 to 26.5]
Statistical Analysis 42: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 42_Week 11, ≥50% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.0006, Chi-squared; Risk Difference (RD) = 17.7, 95% CI 2-sided [7.8 to 27.6]
Statistical Analysis 43: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 43_Week 11, ≥75% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.0075, Chi-squared; Risk Difference (RD) = 15.0, 95% CI 2-sided [4.1 to 25.8]
Statistical Analysis 44: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 44_Week 11, ≥75% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.0010, Chi-squared; Risk Difference (RD) = 18.5, 95% CI 2-sided [7.6 to 29.30]
Statistical Analysis 45: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 45_Week 12, ≥50% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.0001, Chi-squared; Risk Difference (RD) = 20.0, 95% CI 2-sided [10.0 to 29.9]
Statistical Analysis 46: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 46_Week 12, ≥50% reduction, E4 20 mg vs placebo; Test type: Superiority; p < 0.0001, Chi-squared; Risk Difference (RD) = 20.4, 95% CI 2-sided [10.5 to 30.3]
Statistical Analysis 47: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 47_Week 12, ≥75% reduction, E4 15 mg vs placebo; Test type: Superiority; p = 0.0392, Chi-squared; Risk Difference (RD) = 11.7, 95% CI 2-sided [0.7 to 22.7]
Statistical Analysis 48: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 48_Week 12, ≥75% reduction, E4 20 mg vs placebo; Test type: Superiority; p = 0.0007, Chi-squared; Risk Difference (RD) = 19.5, 95% CI 2-sided [8.5 to 30.6]

7. Secondary Outcome: Percentage of Subjects With a Clinically Important Difference (CID) Compared With Baseline in the Weekly Frequency of Moderate to Severe VMS -- Week 4 and Week 12 -- Clinical Global Impression (CGI) Questionnaire -- (Efficacy Study Part)
Description: Percentage of subjects with a clinically important difference (CID) compared with baseline in the weekly frequency of moderate to severe VMS after Week 4 and Week 12, using the Clinical Global Impression (CGI) questionnaire (Efficacy Study Part).
  CGI questionnaire: questionnaire in which subjects were to answer the question "Rate the total improvement, whether or not in your judgement it is due entirely to drug treatment. Compared to your condition at administration to the study, how much has it changed?". The options were: very much improved, much improved, minimally improved, no change, minimally worse, much worse, and very much worse.
  CID (=Clinically Important Difference) = much improved + very much improved; MCID (=Minimally Clinically Important Difference) = minimally improved.
Time Frame: Week 4, Week 12.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
percentage of participants
  Week 4, CID: number analyzed (Participants) | 170 | 175 | 173
  Week 4, CID | 37.6 | 52.6 | 35.8
  Week 4, MCID: number analyzed (Participants) | 170 | 175 | 173
  Week 4, MCID | 46.5 | 29.7 | 37.6
  Week 4, Worsen/No Change: number analyzed (Participants) | 170 | 175 | 173
  Week 4, Worsen/No Change | 15.9 | 17.7 | 26.6
  Week 12, CID: number analyzed (Participants) | 148 | 143 | 144
  Week 12, CID | 63.5 | 71.3 | 52.8
  Week 12, MCID: number analyzed (Participants) | 148 | 143 | 144
  Week 12, MCID | 26.4 | 18.2 | 31.3
  Week 12, Worsen/No Change: number analyzed (Participants) | 148 | 143 | 144
  Week 12, Worsen/No Change | 10.1 | 10.5 | 16.0
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 4, CID, E4 15 mg vs Placebo; Test type: Superiority; p = 0.7283, Chi-squared; Risk Difference (RD) = 1.8, 95% CI 2-sided [-8.4 to 12.0]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 4, CID, E4 20 mg vs Placebo; Test type: Superiority; p = 0.0017, Chi-squared; Risk Difference (RD) = 16.7, 95% CI 2-sided [6.4 to 27.0]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 4, MCID, E4 15 mg vs Placebo; Test type: Superiority; p = 0.0950, Chi-squared; Risk Difference (RD) = 8.9, 95% CI 2-sided [-1.5 to 19.3]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 4, MCID, E4 20 mg vs Placebo; Test type: Superiority; p = 0.1208, Chi-squared; Risk Difference (RD) = -7.9, 95% CI 2-sided [-17.8 to 2.0]
Statistical Analysis 5: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 5_Week 4, Worsen/No change, E4 15 mg vs Placebo; Test type: Superiority; p = 0.0154, Chi-squared; Risk Difference (RD) = -10.7, 95% CI 2-sided [-19.3 to -2.1]
Statistical Analysis 6: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 6_Week 4, Worsen/No change, E4 20 mg vs Placebo; Test type: Superiority; p = 0.0461, Chi-squared; Risk Difference (RD) = -8.9, 95% CI 2-sided [-17.6 to -0.2]
Statistical Analysis 7: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 7_Week 12, CID, E4 15 mg vs Placebo; Test type: Superiority; p = 0.0629, Chi-squared; Risk Difference (RD) = 10.7, 95% CI 2-sided [-0.5 to 22.0]
Statistical Analysis 8: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 8_Week 12, CID, E4 20 mg vs Placebo; Test type: Superiority; p = 0.0012, Chi-squared; Risk Difference (RD) = 18.6, 95% CI 2-sided [7.5 to 29.6]
Statistical Analysis 9: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 9_Week 12, MCID, E4 15 mg vs Placebo; Test type: Superiority; p = 0.3552, Chi-squared; Risk Difference (RD) = -4.9, 95% CI 2-sided [-15.3 to 5.5]
Statistical Analysis 10: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 10_Week 12, MCID, E4 20 mg vs Placebo; Test type: Superiority; p = 0.0103, Chi-squared; Risk Difference (RD) = -13.1, 95% CI 2-sided [-22.9 to -3.2]
Statistical Analysis 11: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 11_Week 12, Worsen/No change, E4 15 mg vs Placebo; Test type: Superiority; p = 0.1383, Chi-squared; Risk Difference (RD) = -5.8, 95% CI 2-sided [-13.5 to 1.9]
Statistical Analysis 12: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 12_Week 12, Worsen/No change, E4 20 mg vs Placebo; Test type: Superiority; p = 0.1706, Chi-squared; Risk Difference (RD) = -5.5, 95% CI 2-sided [-13.3 to 2.3]

8. Secondary Outcome: Total Cholesterol -- (Efficacy Study Part)
Description: Serum concentration of total cholesterol (Efficacy study part).
  Lipid Metabolism: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: Intention-to-treat (ITT) Set: included all subjects who received at least one dose of randomized study medication. All analyses on this set were based on the randomized treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
mmol/L
  Week 12: number analyzed (Participants) | 150 | 144 | 150
  Week 12 | -0.08 [-0.20 to 0.04] | -0.07 [-0.20 to 0.05] | 0.06 [-0.06 to 0.19]
  Week 52: number analyzed (Participants) | 93 | 83 | 102
  Week 52 | -0.25 [-0.40 to -0.10] | -0.26 [-0.41 to -0.10] | -0.02 [-0.16 to 0.13]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.1565, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.15, 95% CI 2-sided [-0.34 to 0.04]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.1823, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.14, 95% CI 2-sided [-0.33 to 0.05]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.0460, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.23, 95% CI 2-sided [-0.46 to -0.00]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.0417, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.24, 95% CI 2-sided [-0.47 to -0.01]

9. Secondary Outcome: Total Cholesterol -- (Safety Study Part)
Description: Serum concentration of total cholesterol (Safety study part).
  Lipid Metabolism: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: Safety analysis set (SAF): included all subjects who received at least one dose of study medication.
  The SAF was used for all analyses of safety and background characteristics.
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Estetrol 20 mg - Safety Study Part
Number analyzed (Participants) | 430
mmol/L
  Week 12: number analyzed (Participants) | 292
  Week 12 | -0.139 [-0.22 to -0.06]
  Week 52: number analyzed (Participants) | 143
  Week 52 | -0.317 [-0.43 to -0.20]

10. Secondary Outcome: Cholesterol/High-density Lipoprotein (HDL) Ratio -- (Efficacy Study Part)
Description: Cholesterol/High-density lipoprotein (HDL) Ratio (Efficacy study part).
  Lipid Metabolism: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Cholesterol/HDL Ratio
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
Cholesterol/HDL Ratio
  Week 12: number analyzed (Participants) | 149 | 144 | 145
  Week 12 | -0.06 [-0.16 to 0.05] | -0.18 [-0.29 to -0.07] | 0.02 [-0.08 to 0.13]
  Week 52: number analyzed (Participants) | 91 | 82 | 98
  Week 52 | -0.11 [-0.24 to 0.02] | -0.08 [-0.22 to 0.05] | 0.01 [-0.11 to 0.13]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.4616, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.08, 95% CI 2-sided [-0.24 to 0.09]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.0112, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.20, 95% CI 2-sided [-0.37 to -0.04]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.2773, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.12, 95% CI 2-sided [-0.32 to 0.07]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.4881, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.09, 95% CI 2-sided [-0.29 to 0.11]

11. Secondary Outcome: Cholesterol/High-density Lipoprotein (HDL) Ratio -- (Safety Study Part).
Description: Cholesterol/High-density lipoprotein (HDL) Ratio (Safety study part).
  Lipid Metabolism: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: Cholesterol/HDL Ratio
Arm/Group | Estetrol 20 mg - Safety Study Part
Number analyzed (Participants) | 430
Cholesterol/HDL Ratio
  Week 12: number analyzed (Participants) | 286
  Week 12 | -0.158 [-0.23 to -0.09]
  Week 52: number analyzed (Participants) | 139
  Week 52 | -0.146 [-0.24 to -0.05]

12. Secondary Outcome: High-density Lipoprotein (HDL)-Cholesterol -- (Efficacy Study Part)
Description: Serum concentration of high-density lipoprotein (HDL)-cholesterol (Efficacy study part).
  Lipid Metabolism: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
mmol/L
  Week 12: number analyzed (Participants) | 149 | 144 | 145
  Week 12 | 0.00 [-0.04 to 0.04] | 0.05 [0.01 to 0.09] | 0.02 [-0.02 to 0.06]
  Week 52: number analyzed (Participants) | 91 | 82 | 98
  Week 52 | -0.02 [-0.07 to 0.03] | -0.03 [-0.08 to 0.02] | -0.01 [-0.06 to 0.04]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.7875, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.02, 95% CI 2-sided [-0.08 to 0.040]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.3092, Linear Mixed Model for Repeated Measures; Least square mean difference = 0.04, 95% CI 2-sided [-0.02 to 0.10]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.9129, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.01, 95% CI 2-sided [-0.08 to 0.06]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.8023, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.02, 95% CI 2-sided [-0.09 to 0.06]

13. Secondary Outcome: High-density Lipoprotein (HDL)-Cholesterol -- (Safety Study Part)
Description: Serum concentration of total HDL cholesterol (Safety study part).
  Lipid Metabolism: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Estetrol 20 mg - Safety Study Part
Number analyzed (Participants) | 430
mmol/L
  Week 12: number analyzed (Participants) | 287
  Week 12 | 0.037 [0.01 to 0.06]
  Week 52: number analyzed (Participants) | 139
  Week 52 | -0.024 [-0.06 to 0.01]

14. Secondary Outcome: Low-density Lipoprotein (LDL)-Cholesterol -- (Efficacy Study Part)
Description: Serum concentration of low-density lipoprotein (LDL)-cholesterol (Efficacy study part)
  Lipid Metabolism: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
mmol/L
  Week 12: number analyzed (Participants) | 150 | 143 | 149
  Week 12 | -0.12 [-0.23 to -0.01] | -0.10 [-0.22 to 0.01] | 0.11 [-0.01 to 0.22]
  Week 52: number analyzed (Participants) | 93 | 82 | 101
  Week 52 | -0.21 [-0.35 to -0.07] | -0.20 [-0.35 to -0.05] | 0.10 [-0.04 to 0.23]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.0084, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.23, 95% CI 2-sided [-0.41 to -0.05]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.0146, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.21, 95% CI 2-sided [-0.39 to -0.04]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.0029, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.30, 95% CI 2-sided [-0.51 to -0.09]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.0045, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.30, 95% CI 2-sided [-0.51 to -0.08]

15. Secondary Outcome: Low-density Lipoprotein (LDL)-Cholesterol -- (Safety Study Part)
Description: Serum Concentration of LDL-cholesterol (Safety study part).
  Lipid Metabolism: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Estetrol 20 mg - Safety Study Part
Number analyzed (Participants) | 430
mmol/L
  Week 12: number analyzed (Participants) | 291
  Week 12 | -0.175 [-0.25 to -0.10]
  Week 52: number analyzed (Participants) | 141
  Week 52 | -0.286 [-0.40 to -0.18]

16. Secondary Outcome: Lipoprotein(a) -- (Efficacy Study Part)
Description: Serum concentration of lipoprotein(a) (Efficacy study part).
  Lipid Metabolism: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
mg/dL
  Week 12: number analyzed (Participants) | 149 | 143 | 151
  Week 12 | -3.35 [-4.84 to -1.85] | -4.04 [-5.54 to -2.53] | -0.01 [-1.48 to 1.47]
  Week 52: number analyzed (Participants) | 90 | 82 | 100
  Week 52 | -2.38 [-4.20 to -0.56] | -2.11 [-4.02 to -0.21] | 0.62 [-1.11 to 2.35]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.0026, Linear Mixed Model for Repeated Measures; Least square mean difference = -3.34, 95% CI 2-sided [-5.63 to -1.05]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.0002, Linear Mixed Model for Repeated Measures; Least square mean difference = -4.03, 95% CI 2-sided [-6.31 to -1.75]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.0295, Linear Mixed Model for Repeated Measures; Least square mean difference = -3.01, 95% CI 2-sided [-5.75 to -0.26]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.0564, Linear Mixed Model for Repeated Measures; Least square mean difference = -2.73, 95% CI 2-sided [-5.53 to 0.06]

17. Secondary Outcome: Lipoprotein(a) -- (Safety Study Part)
Description: Serum Concentration of Lipoprotein(a) (Safety study part).
  Lipid Metabolism: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Estetrol 20 mg - Safety Study Part
Number analyzed (Participants) | 430
mg/dL
  Week 12: number analyzed (Participants) | 287
  Week 12 | -2.20 [-3.66 to -0.73]
  Week 52: number analyzed (Participants) | 140
  Week 52 | -0.81 [-3.08 to 1.46]

18. Secondary Outcome: Triglycerides -- (Efficacy Study Part)
Description: Serum concentration of triglycerides (Efficacy study part).
  Lipid Metabolism: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
mmol/L
  Week 12: number analyzed (Participants) | 150 | 144 | 149
  Week 12 | 0.17 [0.05 to 0.28] | 0.14 [0.03 to 0.26] | -0.07 [-0.19 to 0.04]
  Week 52: number analyzed (Participants) | 93 | 82 | 101
  Week 52 | 0.14 [0.00 to 0.28] | 0.21 [0.06 to 0.35] | 0.00 [-0.13 to 0.13]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.0051, Linear Mixed Model for Repeated Measures; Least square mean difference = 0.24, 95% CI 2-sided [0.06 to 0.42]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.0126, Linear Mixed Model for Repeated Measures; Least square mean difference = 0.22, 95% CI 2-sided [0.04 to 0.40]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.2372, Linear Mixed Model for Repeated Measures; Least square mean difference = 0.14, 95% CI 2-sided [-0.07 to 0.35]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.0644, Linear Mixed Model for Repeated Measures; Least square mean difference = 0.20, 95% CI 2-sided [-0.01 to 0.42]

19. Secondary Outcome: Triglycerides -- (Safety Study Part)
Description: Serum concentration of triglycerides (Safety study part).
  Lipid Metabolism: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: Safety analysis set (SAF): included all subjects who received at least one dose of study drug.
  The SAF was used for all analyses of safety and background characteristics.
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Estetrol 20 mg - Safety Study Part
Number analyzed (Participants) | 430
mmol/L
  Week 12: number analyzed (Participants) | 292
  Week 12 | 0.195 [0.12 to 0.27]
  Week 52: number analyzed (Participants) | 141
  Week 52 | 0.202 [0.07 to 0.34]

20. Secondary Outcome: Hemoglobin A1c -- (Efficacy Study Part)
Description: Hemoglobin A1c (Efficacy study part).
  Glucose metabolism parameters: Change from Baseline to Week 12 and Week 52.
  Hemoglobin A1c = Glycated hemoglobin
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of glycated hemoglobin
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
percentage of glycated hemoglobin
  Week 12: number analyzed (Participants) | 150 | 140 | 147
  Week 12 | -0.02 [-0.07 to 0.04] | -0.09 [-0.14 to -0.03] | 0.02 [-0.03 to 0.07]
  Week 52: number analyzed (Participants) | 92 | 83 | 100
  Week 52 | -0.08 [-0.15 to -0.02] | -0.15 [-0.22 to -0.08] | -0.08 [-0.15 to -0.02]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.5631, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.04, 95% CI 2-sided [-0.12 to 0.05]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.0174, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.11, 95% CI 2-sided [-0.20 to -0.02]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.9992, Linear Mixed Model for Repeated Measures; Least square mean difference = 0.00, 95% CI 2-sided [-0.10 to 0.10]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.2941, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.07, 95% CI 2-sided [-0.17 to 0.04]

21. Secondary Outcome: Hemoglobin A1c -- (Safety Study Part)
Description: Hemoglobin A1c (Safety study part).
  Glucose metabolism parameters: Change from Baseline to Week 12 and Week 52.
  Hemoglobin A1c = Glycated hemoglobin
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of glycated hemoglobin
Arm/Group | Estetrol 20 mg - Safety Study Part
Number analyzed (Participants) | 430
percentage of glycated hemoglobin
  Week 12: number analyzed (Participants) | 285
  Week 12 | -0.05 [-0.07 to -0.02]
  Week 52: number analyzed (Participants) | 138
  Week 52 | -0.02 [-0.08 to 0.04]

22. Secondary Outcome: Fasting Glucose -- (Efficacy Study Part)
Description: Concentration of fasting glucose in plasma.
  Glucose metabolism parameters: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
mmol/L
  Week 12: number analyzed (Participants) | 150 | 137 | 138
  Week 12 | 0.01 [-0.11 to 0.12] | -0.04 [-0.15 to 0.08] | 0.06 [-0.05 to 0.18]
  Week 52: number analyzed (Participants) | 88 | 81 | 98
  Week 52 | -0.04 [-0.19 to 0.10] | 0.00 [-0.15 to 0.15] | -0.04 [-0.17 to 0.10]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.7112, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.06, 95% CI 2-sided [-0.24 to 0.12]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.3618, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.10, 95% CI 2-sided [-0.28 to 0.08]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.9933, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.01, 95% CI 2-sided [-0.23 to 0.21]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.9024, Linear Mixed Model for Repeated Measures; Least square mean difference = 0.099, 95% CI 2-sided [-0.18 to 0.26]

23. Secondary Outcome: Fasting Glucose -- (Safety Study Part)
Description: Concentration of fasting glucose in plasma.
  Glucose metabolism parameters: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Estetrol 20 mg - Safety Study Part
Number analyzed (Participants) | 430
mmol/L
  Week 12: number analyzed (Participants) | 277
  Week 12 | 0.074 [-0.02 to 0.17]
  Week 52: number analyzed (Participants) | 139
  Week 52 | 0.092 [-0.08 to 0.27]

24. Secondary Outcome: Insulin Resistance (HOMA-IR) -- Homeostasis Model Assessment -- (Efficacy Study Part)
Description: Insulin resistance (HOMA-IR) -- Homeostasis model assessment (Efficacy study part).
  Glucose Metabolism parameters: Change from Baseline to Week 12 and Week 52.
  HOMA-IR is a mathematical homeostasis model assessment (HOMA) that evaluates systemic insulin resistance (IR).
  The HOMA-IR score is calculated as the product of fasting insulin and fasting glucose values divided by a constant. Low HOMA-IR means that a small amount of the hormone insulin is sufficient to keep blood sugars in good balance.
  HOMA-IR values less than 1.0 mean insulin-sensitivity which is optimal. Values ≥1.9 are indicative of early insulin resistance, and ≥2.9 indicate significant insulin resistance.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: index
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
index
  Week 12: number analyzed (Participants) | 141 | 133 | 138
  Week 12 | -0.09 [-0.66 to 0.49] | -0.02 [-0.62 to 0.57] | 0.07 [-0.51 to 0.65]
  Week 52: number analyzed (Participants) | 80 | 73 | 94
  Week 52 | -0.66 [-1.42 to 0.09] | 0.27 [-0.53 to 1.07] | -0.46 [-1.16 to 0.24]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.8961, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.16, 95% CI 2-sided [-1.05 to 0.74]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.9619, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.09, 95% CI 2-sided [-0.99 to 0.81]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.8920, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.20, 95% CI 2-sided [-1.33 to 0.92]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.2826, Linear Mixed Model for Repeated Measures; Least square mean difference = 0.73, 95% CI 2-sided [-0.43 to 1.89]

25. Secondary Outcome: Insulin Resistance (HOMA-IR) -- Homeostasis Model Assessment -- (Safety Study Part)
Description: Insulin resistance (HOMA-IR) -- Homeostasis model assessment (Safety study part).
  Glucose Metabolism parameters: Change from Baseline to Week 12 and Week 52.
  HOMA-IR is a mathematical homeostasis model assessment (HOMA) that evaluates systemic insulin resistance (IR).
  The HOMA-IR score is calculated as the product of fasting insulin and fasting glucose values divided by a constant. Low HOMA-IR means that a small amount of the hormone insulin is sufficient to keep blood sugars in good balance.
  HOMA-IR values less than 1.0 mean insulin-sensitivity which is optimal. Values ≥1.9 are indicative of early insulin resistance, and ≥2.9 indicate significant insulin resistance.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 19
Measure: Mean (95% Confidence Interval); unit: index
Arm/Group | Estetrol 20 mg - Safety Study Part
Number analyzed (Participants) | 430
index
  Week 12: number analyzed (Participants) | 276
  Week 12 | 0.124 [-0.33 to 0.58]
  Week 52: number analyzed (Participants) | 132
  Week 52 | -0.156 [-0.76 to 0.45]

26. Secondary Outcome: Insulin -- (Efficacy Study Part)
Description: Serum concentration of insulin (Efficacy study part).
  Glucose metabolism parameters: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
pmol/L
  Week 12: number analyzed (Participants) | 144 | 139 | 144
  Week 12 | -4.28 [-19.18 to 10.62] | -2.66 [-17.67 to 12.36] | -0.41 [-15.18 to 14.36]
  Week 52: number analyzed (Participants) | 83 | 75 | 96
  Week 52 | -16.40 [-35.57 to 2.78] | 6.48 [-13.92 to 26.89] | -10.67 [-28.54 to 7.21]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.9039, Linear Mixed Model for Repeated Measures; Least square mean difference = -3.87, 95% CI 2-sided [-26.86 to 19.12]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.9660, Linear Mixed Model for Repeated Measures; Least square mean difference = -2.24, 95% CI 2-sided [-25.12 to 20.63]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.8708, Linear Mixed Model for Repeated Measures; Least square mean difference = -5.73, 95% CI 2-sided [-34.55 to 23.08]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.3357, Linear Mixed Model for Repeated Measures; Least square mean difference = 17.15, 95% CI 2-sided [-12.48 to 46.77]

27. Secondary Outcome: Insulin -- (Safety Study Part)
Description: Serum concentration of insulin (Safety study part).
  Glucose metabolism parameters: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 19
Measure: Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Estetrol 20 mg - Safety Study Part
Number analyzed (Participants) | 430
pmol/L
  Week 12: number analyzed (Participants) | 279
  Week 12 | 1.2 [-9.44 to 11.89]
  Week 52: number analyzed (Participants) | 134
  Week 52 | -5.2 [-19.98 to 9.65]

28. Secondary Outcome: Angiotensinogen -- (Efficacy Study Part)
Description: Angiotensinogen (Efficacy study part).
  Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
µg/mL
  Week 12: number analyzed (Participants) | 135 | 131 | 143
  Week 12 | 16.86 [13.93 to 19.80] | 18.90 [15.95 to 21.84] | -0.50 [-3.31 to 2.31]
  Week 52: number analyzed (Participants) | 87 | 73 | 94
  Week 52 | 18.47 [15.01 to 21.93] | 21.22 [17.39 to 25.04] | 1.03 [-2.25 to 4.30]
Statistical Analysis 1: Comparison: Placebo - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures; Least square mean difference = 17.36, 95% CI 2-sided [12.76 to 21.96]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures; Least square mean difference = 19.39, 95% CI 2-sided [14.80 to 23.98]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures; Least square mean difference = 17.44, 95% CI 2-sided [12.05 to 22.83]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures; Least square mean difference = 20.19, 95% CI 2-sided [14.50 to 25.89]

29. Secondary Outcome: Antithrombin Activity (AT III) -- (Efficacy Study Part)
Description: Antithrombin Activity (AT III) -- (Efficacy study part)
  Hemostasis parameters: Change from Baseline to Week 12 and Week 52.
  Antithrombin Activity (AT III) is a key biomarker that measures how effectively antithrombin, a natural anticoagulant protein, functions in the blood.
  The functional AT III assay is based on the principle of inhibition of Factor Xa by antithrombin in the presence of heparin.
  Antithrombin Activity results are expressed as a percentage, with normal levels ranging between 80% and 120%. Lower than normal levels may indicate an increased risk of blood clotting disorders, while elevated levels can occur during inflammation or certain physiological conditions.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of activity
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
percentage of activity
  Week 12: number analyzed (Participants) | 137 | 137 | 144
  Week 12 | -8.99 [-11.23 to -6.75] | -8.97 [-11.28 to -6.65] | -0.71 [-2.96 to 1.52]
  Week 52: number analyzed (Participants) | 86 | 74 | 94
  Week 52 | -7.66 [-10.43 to -4.88] | -5.49 [-8.63 to -2.35] | 0.02 [-2.69 to 2.73]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p < 0.0001, Linear Mixed Model for Repeated Measures; Least square mean difference = -8.28, 95% CI 2-sided [-11.86 to -4.70]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p < 0.0001, Linear Mixed Model for Repeated Measures; Least square mean difference = -8.25, 95% CI 2-sided [-11.90 to -4.61]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.0002, Linear Mixed Model for Repeated Measures; Least square mean difference = -7.68, 95% CI 2-sided [-12.07 to -3.29]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.0181, Linear Mixed Model for Repeated Measures; Least square mean difference = -5.51, 95% CI 2-sided [-10.21 to -0.82]

30. Secondary Outcome: Activated Partial Thromboplastin Time (aPTT) Based Activated Protein-C Resistance (APCr) (APCR-V Ratio) -- (Efficacy Study Part)
Description: Activated partial thromboplastin time (aPTT) based activated Protein-C resistance (APCr) (APCR-V ratio) (Efficacy study part).
  Hemostasis parameters: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: APCR-V ratio
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
APCR-V ratio
  Week 12: number analyzed (Participants) | 137 | 137 | 144
  Week 12 | 0.04 [-0.00 to 0.08] | 0.02 [-0.02 to 0.07] | 0.05 [0.01 to 0.09]
  Week 52: number analyzed (Participants) | 86 | 74 | 93
  Week 52 | 0.08 [0.03 to 0.13] | 0.05 [-0.00 to 0.11] | 0.09 [0.04 to 0.13]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.8862, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.01, 95% CI 2-sided [-0.08 to 0.05]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.6013, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.02, 95% CI 2-sided [-0.09 to 0.04]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.9723, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.01, 95% CI 2-sided [-0.08 to 0.07]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.5778, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.03, 95% CI 2-sided [-0.11 to 0.05]

31. Secondary Outcome: Prothrombin Fragment 1 + 2 -- (Efficacy Study Part)
Description: Prothrombin fragment 1 + 2 (Efficacy study part).
  Hemostasis parameters: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
pmol/L
  Week 12: number analyzed (Participants) | 139 | 135 | 144
  Week 12 | -44.61 [-104.50 to 15.27] | -57.53 [-120.31 to 5.25] | -50.48 [-110.13 to 9.18]
  Week 52: number analyzed (Participants) | 86 | 73 | 94
  Week 52 | -69.85 [-146.81 to 7.11] | -95.03 [-183.39 to 6.66] | -23.39 [-97.76 to 50.99]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.9865, Linear Mixed Model for Repeated Measures; Least square mean difference = 5.86, 95% CI 2-sided [-89.50 to 101.23]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.9814, Linear Mixed Model for Repeated Measures; Least square mean difference = -7.05, 95% CI 2-sided [-104.73 to 90.63]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.6049, Linear Mixed Model for Repeated Measures; Least square mean difference = -46.46, 95% CI 2-sided [-167.23 to 74.30]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.3717, Linear Mixed Model for Repeated Measures; Least square mean difference = -71.64, 95% CI 2-sided [-202.08 to 58.81]

32. Secondary Outcome: Factor VIII -- (Efficacy Study Part)
Description: Factor VIII (Efficacy study part).
  Hemostasis parameters: Change from Baseline to Week 12 and Week 52.
  This test measures the activity of Factor VIII which is an essential protein for effective formation of a blood clot.
  Factor VIII activity results are expressed as a percentage, with normal levels ranging from 50% to 150%. Lower than normal levels can indicate bleeding disorders such as hemophilia A or acquired Factor VIII deficiency.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of activity
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
percentage of activity
  Week 12: number analyzed (Participants) | 137 | 137 | 145
  Week 12 | -0.52 [-6.07 to 5.02] | 3.21 [-2.49 to 8.92] | -2.45 [-7.94 to 3.04]
  Week 52: number analyzed (Participants) | 86 | 74 | 93
  Week 52 | -2.39 [-9.13 to 4.35] | 6.99 [-0.57 to 14.55] | 1.47 [-5.13 to 8.07]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.8439, Linear Mixed Model for Repeated Measures; Least square mean difference = 1.93, 95% CI 2-sided [-6.89 to 10.74]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.2727, Linear Mixed Model for Repeated Measures; Least square mean difference = 5.66, 95% CI 2-sided [-3.28 to 14.61]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.6389, Linear Mixed Model for Repeated Measures; Least square mean difference = -3.86, 95% CI 2-sided [-14.53 to 6.81]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.4544, Linear Mixed Model for Repeated Measures; Least square mean difference = 5.52, 95% CI 2-sided [-5.84 to 16.88]

33. Secondary Outcome: Endogenous Thrombin Potential (ETP)-Based Activated Protein-C Sensitivity Ratio (APCsr ETP) -- (Efficacy Study Part)
Description: Endogenous thrombin potential (ETP)-based activated Protein-C sensitivity ratio (APCsr ETP) (Efficacy study part).
  Hemostasis parameters: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: APCsr ETP ratio
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
APCsr ETP ratio
  Week 12: number analyzed (Participants) | 126 | 126 | 138
  Week 12 | 0.65 [0.36 to 0.94] | 0.84 [0.57 to 1.12] | 0.08 [-0.19 to 0.35]
  Week 52: number analyzed (Participants) | 80 | 71 | 87
  Week 52 | 0.66 [0.32 to 1.00] | 0.90 [0.55 to 1.26] | 0.47 [0.15 to 0.78]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.0084, Linear Mixed Model for Repeated Measures; Least square mean difference = 0.57, 95% CI 2-sided [0.13 to 1.02]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.0002, Linear Mixed Model for Repeated Measures; Least square mean difference = 0.77, 95% CI 2-sided [0.33 to 1.20]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.6337, Linear Mixed Model for Repeated Measures; Least square mean difference = 0.19, 95% CI 2-sided [-0.33 to 0.72]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.1287, Linear Mixed Model for Repeated Measures; Least square mean difference = 0.44, 95% CI 2-sided [-0.10 to 0.98]

34. Secondary Outcome: Protein-C -- (Efficacy Study Part)
Description: Protein-C (Efficacy study part).
  Hemostasis parameters: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of activity
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
percentage of activity
  Week 12: number analyzed (Participants) | 137 | 137 | 145
  Week 12 | -4.82 [-7.53 to -2.11] | -2.34 [-5.12 to 0.44] | -2.37 [-5.05 to 0.31]
  Week 52: number analyzed (Participants) | 86 | 74 | 94
  Week 52 | -6.13 [-9.38 to -2.89] | -3.93 [-7.55 to -0.32] | -3.76 [-6.93 to -0.59]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.3445, Linear Mixed Model for Repeated Measures; Least square mean difference = -2.45, 95% CI 2-sided [-6.76 to 1.86]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.9998, Linear Mixed Model for Repeated Measures; Least square mean difference = 0.03, 95% CI 2-sided [-4.33 to 4.40]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.4874, Linear Mixed Model for Repeated Measures; Least square mean difference = -2.38, 95% CI 2-sided [-7.51 to 2.76]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.9964, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.17, 95% CI 2-sided [-5.61 to 5.26]

35. Secondary Outcome: Free Protein-S -- (Efficacy Study Part)
Description: Free Protein-S (Efficacy study part).
  Hemostasis parameters: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: percent free protein S
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
percent free protein S
  Week 12: number analyzed (Participants) | 137 | 137 | 145
  Week 12 | -4.96 [-7.04 to -2.87] | -5.79 [-7.86 to -3.71] | -1.01 [-3.05 to 1.02]
  Week 52: number analyzed (Participants) | 86 | 74 | 94
  Week 52 | -4.84 [-7.41 to -2.26] | -4.06 [-6.84 to -1.28] | -0.28 [-2.74 to 2.19]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.0119, Linear Mixed Model for Repeated Measures; Least square mean difference = -3.94, 95% CI 2-sided [-7.12 to -0.76]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.0017, Linear Mixed Model for Repeated Measures; Least square mean difference = -4.77, 95% CI 2-sided [-7.93 to -1.62]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.0186, Linear Mixed Model for Repeated Measures; Least square mean difference = -4.56, 95% CI 2-sided [-8.46 to -0.66]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.0687, Linear Mixed Model for Repeated Measures; Least square mean difference = -3.79, 95% CI 2-sided [-7.81 to 0.24]

36. Secondary Outcome: Sex Hormone Binding Globulin (SHBG) -- (Efficacy Study Part)
Description: Sex Hormone Binding Globulin (SHBG) (Efficacy study part).
  Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
nmol/L
  Week 12: number analyzed (Participants) | 137 | 134 | 144
  Week 12 | 26.76 [19.37 to 34.15] | 43.85 [36.53 to 51.17] | -1.14 [-8.15 to 5.87]
  Week 52: number analyzed (Participants) | 88 | 75 | 95
  Week 52 | 31.47 [23.26 to 39.69] | 50.70 [41.99 to 59.42] | 1.55 [-6.23 to 9.34]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures; Least square mean difference = 27.90, 95% CI 2-sided [16.40 to 39.41]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures; Least square mean difference = 44.99, 95% CI 2-sided [33.53 to 56.44]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures; Least square mean difference = 29.92, 95% CI 2-sided [17.13 to 42.71]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures; Least square mean difference = 49.15, 95% CI 2-sided [35.92 to 62.37]

37. Secondary Outcome: Calcium -- (Efficacy Study Part)
Description: Calcium (Efficacy study part).
  Bone turnover markers: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
mmol/L
  Week 12: number analyzed (Participants) | 150 | 143 | 150
  Week 12 | -0.04 [-0.06 to -0.03] | -0.08 [-0.09 to -0.06] | 0.00 [-0.02 to 0.02]
  Week 52: number analyzed (Participants) | 93 | 83 | 102
  Week 52 | -0.07 [-0.09 to -0.04] | -0.11 [-0.13 to -0.08] | -0.04 [-0.06 to -0.02]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.0004, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.04, 95% CI 2-sided [-0.07 to -0.02]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p < 0.0001, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.08, 95% CI 2-sided [-0.10 to -0.05]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.0898, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.03, 95% CI 2-sided [-0.06 to 0.00]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p < 0.0001, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.07, 95% CI 2-sided [-0.10 to -0.04]

38. Secondary Outcome: C-Terminal Telopeptide Type 1 (CTX-1) -- (Efficacy Study Part)
Description: C-terminal telopeptide type 1 (CTX-1) (Efficacy study part).
  Bone turnover markers: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: µg/L
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
µg/L
  Week 12: number analyzed (Participants) | 140 | 135 | 143
  Week 12 | -0.15 [-0.18 to -0.12] | -0.15 [-0.19 to -0.12] | -0.02 [-0.05 to 0.01]
  Week 52: number analyzed (Participants) | 84 | 73 | 95
  Week 52 | -0.19 [-0.22 to -0.15] | -0.16 [-0.20 to -0.12] | -0.02 [-0.05 to 0.02]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p < 0.0001, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.13, 95% CI 2-sided [-0.18 to -0.08]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p < 0.0001, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.14, 95% CI 2-sided [-0.18 to -0.09]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p < 0.0001, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.17, 95% CI 2-sided [-0.23 to -0.11]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p < 0.0001, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.14, 95% CI 2-sided [-0.20 to -0.08]

39. Secondary Outcome: Procollagen I N-Terminal Propeptide (PINP) -- (Efficacy Study Part)
Description: Procollagen I N-Terminal Propeptide (PINP) (Efficacy study part).
  Bone turnover markers: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: µg/L
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
µg/L
  Week 12: number analyzed (Participants) | 141 | 135 | 143
  Week 12 | -8.45 [-11.99 to -4.91] | -13.84 [-17.40 to -10.27] | -2.22 [-5.71 to 1.26]
  Week 52: number analyzed (Participants) | 82 | 72 | 95
  Week 52 | -16.08 [-20.57 to -11.59] | -13.83 [-18.63 to -9.03] | -0.15 [-4.34 to 4.04]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.0220, Linear Mixed Model for Repeated Measures; Least square mean difference = -6.22, 95% CI 2-sided [-11.67 to -0.78]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p < 0.0001, Linear Mixed Model for Repeated Measures; Least square mean difference = -11.61, 95% CI 2-sided [-17.02 to -6.21]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p < 0.0001, Linear Mixed Model for Repeated Measures; Least square mean difference = -15.93, 95% CI 2-sided [-22.70 to -9.17]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p < 0.0001, Linear Mixed Model for Repeated Measures; Least square mean difference = -13.68, 95% CI 2-sided [-20.63 to -6.74]

40. Secondary Outcome: 25-Hydroxyvitamin D -- (Efficacy Study Part)
Description: 25-Hydroxyvitamin D (Efficacy study part).
  Bone turnover markers: Change from Baseline to Week 12 and Week 52.
Time Frame: Day 1 (Baseline), Weeks 12 and 52.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
nmol/L
  Week 12: number analyzed (Participants) | 141 | 138 | 147
  Week 12 | 2.37 [-1.92 to 6.66] | -2.19 [-6.46 to 2.07] | 0.51 [-3.66 to 4.67]
  Week 52: number analyzed (Participants) | 87 | 77 | 97
  Week 52 | 13.89 [8.44 to 19.33] | 5.52 [-0.29 to 11.34] | 7.07 [1.97 to 12.17]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 12 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.7531, Linear Mixed Model for Repeated Measures; Least square mean difference = 1.86, 95% CI 2-sided [-4.69 to 8.42]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 12 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.5548, Linear Mixed Model for Repeated Measures; Least square mean difference = -2.70, 95% CI 2-sided [-9.18 to 3.79]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 52 Estetrol 15 mg vs Placebo; Test type: Superiority; p = 0.1170, Linear Mixed Model for Repeated Measures; Least square mean difference = 6.81, 95% CI 2-sided [-1.36 to 14.99]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52 Estetrol 20 mg vs Placebo; Test type: Superiority; p = 0.8885, Linear Mixed Model for Repeated Measures; Least square mean difference = -1.55, 95% CI 2-sided [-9.97 to 6.87]

41. Secondary Outcome: Health-related Quality of Life (HRQoL) Assessment, Change From Baseline -- Menopause-specific Quality of Life (MENQOL) Questionnaire -- (Efficacy Study Part)
Description: Change from Baseline to W12 and W52 in HRQoL using the MENQOL questionnaire. MENQOL questionnaire=29-item assessment of QoL to capture self-reported information on the presence and bother of symptoms and feelings in the domains of vasomotor, psychosocial, physical and sexual functioning, among midlife women in the immediate post-menopause time.
  For each item, women are asked if they experience that symptom or feeling, and if yes, to rate bother on a scale of 0-6 corresponding to "not at all bothered" to "extremely bothered". Non-endorsement of an item is scored a "1" and endorsement a "2", plus the number of the particular rating, so that the possible score on any item ranges from 1 (not experiencing symptom or feeling) to 8 (extremely bothered).
  Domain score=mean of the item scores in that domain. Total MENQOL=mean of the domain-specific scores. Administered at Day 1 (=day of randomization) for baseline, W12 and W52. It refers to the symptoms experienced over the past month.
Time Frame: Day 1 (Baseline), Week 12, and 52.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part
Number analyzed (Participants) | 192 | 193 | 194
scores on a scale
  Week 12 -- Vasomotor Domain: number analyzed (Participants) | 151 | 145 | 150
  Week 12 -- Vasomotor Domain | -2.83 [-3.15 to -2.51] | -3.15 [-3.48 to -2.83] | -2.38 [-2.70 to -2.06]
  Week 52 -- Vasomotor Domain: number analyzed (Participants) | 93 | 81 | 106
  Week 52 -- Vasomotor Domain | -3.75 [-4.14 to -3.36] | -3.74 [-4.16 to -3.32] | -2.99 [-3.36 to -2.63]
  Week 12 -- Psychosocial Domain: number analyzed (Participants) | 151 | 145 | 150
  Week 12 -- Psychosocial Domain | -1.27 [-1.49 to -1.05] | -1.31 [-1.53 to -1.09] | -1.15 [-1.36 to -0.93]
  Week 52 -- Psychosocial Domain: number analyzed (Participants) | 93 | 81 | 106
  Week 52 -- Psychosocial Domain | -1.57 [-1.83 to -1.30] | -1.17 [-1.45 to -0.89] | -1.25 [-1.50 to -1.00]
  Week 12 -- Physical Domain: number analyzed (Participants) | 151 | 145 | 150
  Week 12 -- Physical Domain | -1.23 [-1.44 to -1.02] | -1.03 [-1.24 to -0.82] | -1.15 [-1.36 to -0.94]
  Week 52 -- Physical Domain: number analyzed (Participants) | 93 | 81 | 106
  Week 52 -- Physical Domain | -1.39 [-1.64 to -1.14] | -1.05 [-1.32 to -0.78] | -1.14 [-1.38 to -0.90]
  Week 12 -- Sexual functioning Domain: number analyzed (Participants) | 151 | 145 | 150
  Week 12 -- Sexual functioning Domain | -1.42 [-1.73 to -1.12] | -1.37 [-1.68 to -1.06] | -1.15 [-1.45 to -0.84]
  Week 52 -- Sexual functioning Domain: number analyzed (Participants) | 93 | 81 | 106
  Week 52 -- Sexual functioning Domain | -1.65 [-2.02 to -1.27] | -1.11 [-1.51 to -0.71] | -1.25 [-1.61 to -0.90]
  Week 12 -- Total MENQOL: number analyzed (Participants) | 151 | 145 | 150
  Week 12 -- Total MENQOL | -1.69 [-1.89 to -1.49] | -1.72 [-1.93 to -1.52] | -1.47 [-1.67 to -1.27]
  Week 52 -- Total MENQOL: number analyzed (Participants) | 93 | 81 | 106
  Week 52 -- Total MENQOL | -2.08 [-2.32 to -1.85] | -1.78 [-2.04 to -1.53] | -1.66 [-1.89 to -1.43]
Statistical Analysis 1: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 1_Week 12, Vasomotor Domain, E4 15 mg vs Placebo; Test type: Superiority; p = 0.0781, Mixed Model for Repeated Measures; Least square mean difference = -0.45, 95% CI 2-sided [-0.95 to 0.04]
Statistical Analysis 2: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 2_Week 12, Vasomotor Domain, E4 20 mg vs Placebo; Test type: Superiority; p = 0.0011, Mixed Model for Repeated Measures; Least square mean difference = -0.78, 95% CI 2-sided [-1.27 to -0.28]
Statistical Analysis 3: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 3_Week 52, Vasomotor Domain, E4 15 mg vs Placebo; Test type: Superiority; p = 0.0085, Linear Mixed Model for Repeated Measures; Least square mean difference = -0.76, 95% CI 2-sided [-1.35 to -0.17]
Statistical Analysis 4: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 4_Week 52, Vasomotor Domain, E4 20 mg vs Placebo; Test type: Superiority; p = 0.0127, Mixed Model for Repeated Measures; Least square mean difference = -0.75, 95% CI 2-sided [-1.35 to -0.14]
Statistical Analysis 5: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 5_Week 12, Psychosocial Domain, E4 15 mg vs Placebo; Test type: Superiority; p = 0.6211, Mixed Model for Repeated Measures; Least square mean difference = -0.12, 95% CI 2-sided [-0.46 to 0.21]
Statistical Analysis 6: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 6_Week 12, Psychosocial Domain, E4 20 mg vs Placebo; Test type: Superiority; p = 0.4544, Mixed Model for Repeated Measures; Least square mean difference = -0.16, 95% CI 2-sided [-0.50 to 0.17]
Statistical Analysis 7: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 7_Week 52, Psychosocial Domain, E4 15 mg vs Placebo; Test type: Superiority; p = 0.1349, Mixed Model for Repeated Measures; Least square mean difference = -0.32, 95% CI 2-sided [-0.72 to 0.08]
Statistical Analysis 8: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 8_Week 52, Psychosocial Domain, E4 20 mg vs Placebo; Test type: Superiority; p = 0.8875, Mixed Model for Repeated Measures; Least square mean difference = 0.08, 95% CI 2-sided [-0.33 to 0.49]
Statistical Analysis 9: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 9_Week 12, Physical Domain, E4 15 mg vs Placebo; Test type: Superiority; p = 0.8109, Mixed Model for Repeated Measures; Least square mean difference = -0.08, 95% CI 2-sided [-0.40 to 0.24]
Statistical Analysis 10: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 10_Week 12, Physical Domain, E4 20 mg vs Placebo; Test type: Superiority; p = 0.6184, Mixed Model for Repeated Measures; Least square mean difference = 0.12, 95% CI 2-sided [-0.20 to 0.44]
Statistical Analysis 11: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 11_Week 52, Physical Domain, E4 15 mg vs Placebo; Test type: Superiority; p = 0.2548, Mixed Model for Repeated Measures; Least square mean difference = -0.25, 95% CI 2-sided [-0.63 to 0.13]
Statistical Analysis 12: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 12_Week 52, Physical Domain, E4 20 mg vs Placebo; Test type: Superiority; p = 0.8282, Mixed Model for Repeated Measures; Least square mean difference = 0.09, 95% CI 2-sided [-0.30 to 0.48]
Statistical Analysis 13: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 13_Week 12, Sexual Domain, E4 15 mg vs Placebo; Test type: Superiority; p = 0.3299, Mixed Model for Repeated Measures; Least square mean difference = -0.27, 95% CI 2-sided [-0.75 to 0.20]
Statistical Analysis 14: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 14_Week 12, Sexual Domain, E4 20 mg vs Placebo; Test type: Superiority; p = 0.4800, Mixed Model for Repeated Measures; Least square mean difference = -0.22, 95% CI 2-sided [-0.69 to 0.25]
Statistical Analysis 15: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 15_Week 52, Sexual Domain, E4 15 mg vs Placebo; Test type: Superiority; p = 0.2133, Mixed Model for Repeated Measures; Least square mean difference = -0.39, 95% CI 2-sided [-0.96 to 0.17]
Statistical Analysis 16: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 16_Week 52, Sexual Domain, E4 20 mg vs Placebo; Test type: Superiority; p = 0.8116, Mixed Model for Repeated Measures; Least square mean difference = 0.14, 95% CI 2-sided [-0.44 to 0.73]
Statistical Analysis 17: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 17_Week 12, Total MENQOL, E4 15 mg vs Placebo; Test type: Superiority; p = 0.1853, Mixed Model for Repeated Measures; Least square mean difference = -0.23, 95% CI 2-sided [-0.53 to 0.08]
Statistical Analysis 18: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 18_Week 12, Total MENQOL, E4 20 mg vs Placebo; Test type: Superiority; p = 0.1176, Mixed Model for Repeated Measures; Least square mean difference = -0.26, 95% CI 2-sided [-0.57 to 0.05]
Statistical Analysis 19: Comparison: Estetrol 15 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 19_Week 52, Total MENQOL, E4 15 mg vs Placebo; Test type: Superiority; p = 0.0176, Mixed Model for Repeated Measures; Least square mean difference = -0.43, 95% CI 2-sided [-0.79 to -0.06]
Statistical Analysis 20: Comparison: Estetrol 20 mg - Efficacy Study Part vs Placebo - Efficacy Study Part; 20_Week 52, Total MENQOL, E4 20 mg vs Placebo; Test type: Superiority; p = 0.6909, Mixed Model for Repeated Measures; Least square mean difference = -0.12, 95% CI 2-sided [-0.49 to 0.25]

42. Secondary Outcome: Health-related Quality of Life (HRQoL) Assessment, Change From Baseline -- Menopause-specific Quality of Life (MENQOL) Questionnaire -- (Safety Study Part)
Description: as for outcome 41
Time Frame: Day 1 (Baseline), Week 12 and 52.
Population: Safety analysis set (SAF): included all subjects who received at least one dose of study medication.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Estetrol 20 mg - Safety Study Part
Number analyzed (Participants) | 430
scores on a scale
  Week 12 -- Vasomotor Domain: number analyzed (Participants) | 290
  Week 12 -- Vasomotor Domain | -3.34 [-3.58 to -3.11]
  Week 52 -- Vasomotor Domain: number analyzed (Participants) | 142
  Week 52 -- Vasomotor Domain | -3.19 [-3.56 to -2.83]
  Week 12 -- Psychosocial Domain: number analyzed (Participants) | 290
  Week 12 -- Psychosocial Domain | -1.20 [-1.40 to -1.01]
  Week 52 -- Psychosocial Domain: number analyzed (Participants) | 142
  Week 52 -- Psychosocial Domain | -1.25 [-1.52 to -0.97]
  Week 12 -- Physical Domain: number analyzed (Participants) | 290
  Week 12 -- Physical Domain | -1.27 [-1.44 to -1.09]
  Week 52 -- Physical Domain: number analyzed (Participants) | 142
  Week 52 -- Physical Domain | -1.11 [-1.37 to -0.86]
  Week 12 -- Sexual functioning Domain: number analyzed (Participants) | 290
  Week 12 -- Sexual functioning Domain | -1.63 [-1.88 to -1.39]
  Week 52 -- Sexual functioning Domain: number analyzed (Participants) | 142
  Week 52 -- Sexual functioning Domain | -1.55 [-1.94 to -1.17]
  Week 12 -- Total MENQOL: number analyzed (Participants) | 290
  Week 12 -- Total MENQOL | -1.86 [-2.01 to -1.71]
  Week 52 -- Total MENQOL: number analyzed (Participants) | 142
  Week 52 -- Total MENQOL | -1.78 [-2.02 to -1.53]

43. Secondary Outcome: Total Score in Treatment Satisfaction (TS) Using the Clinical Global Impression (CGI) Questionnaire -- (Efficacy Study Part, Safety Study Part)
Description: Total score in treatment satisfaction (TS) using the Clinical Global Impression (CGI) questionnaire (Efficacy study part and Safety study part).
  CGI questionnaire: questionnaire in which subjects were to answer the question "Rate the total improvement, whether or not in your judgement it is due entirely to drug treatment. Compared to your condition at administration to the study, how much has it changed?". The options were: very much improved, much improved, minimally improved, no change, minimally worse, much worse, and very much worse.
  Results are shown as percentage of participants.
  TS=Treatment satisfaction
Time Frame: Weeks 4, 12, and 52.
Population: Intention-to-treat (ITT) Set for Efficacy Study Part: included all subjects who received at least one dose of randomized study medication.
  The ITT set was the primary analysis set for the efficacy analyses and all analyses on this set were based on the randomized treatment.
  Safety analysis set (SAF) for Safety Study Part: included all subjects who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part | Estetrol 20 mg - Safety Study Part
Number analyzed (Participants) | 192 | 193 | 194 | 430
percentage of participants
  1_Week 4 - Very Much Improved: number analyzed (Participants) | 173 | 177 | 175 | 374
  1_Week 4 - Very Much Improved | 11.6 | 17.5 | 10.3 | 22.5
  2_Week 4 - Much Improved: number analyzed (Participants) | 173 | 177 | 175 | 374
  2_Week 4 - Much Improved | 25.4 | 34.5 | 25.1 | 36.6
  3_Week 4 - Minimally Improved: number analyzed (Participants) | 173 | 177 | 175 | 374
  3_Week 4 - Minimally Improved | 46.8 | 29.9 | 37.7 | 28.6
  4_Week 4 - No change: number analyzed (Participants) | 173 | 177 | 175 | 374
  4_Week 4 - No change | 14.5 | 16.4 | 24.6 | 10.2
  5_Week 4 - Minimally worse: number analyzed (Participants) | 173 | 177 | 175 | 374
  5_Week 4 - Minimally worse | 0.6 | 0.6 | 1.7 | 1.6
  6_Week 4 - Much worse: number analyzed (Participants) | 173 | 177 | 175 | 374
  6_Week 4 - Much worse | 0.6 | 1.1 | 0.6 | 0.5
  7_Week 4 - Very Much Worse: number analyzed (Participants) | 173 | 177 | 175 | 374
  7_Week 4 - Very Much Worse | 0.6 | 0 | 0 | 0.0
  1_Week 12 - Very Much Improved: number analyzed (Participants) | 151 | 144 | 151 | 285
  1_Week 12 - Very Much Improved | 19.9 | 26.4 | 15.9 | 29.8
  2_Week 12 - Much Improved: number analyzed (Participants) | 151 | 144 | 151 | 285
  2_Week 12 - Much Improved | 43.7 | 45.1 | 37.1 | 44.6
  3_Week 12 - Minimally Improved: number analyzed (Participants) | 151 | 144 | 151 | 285
  3_Week 12 - Minimally Improved | 26.5 | 18.1 | 31.8 | 18.6
  4_Week 12 - No change: number analyzed (Participants) | 151 | 144 | 151 | 285
  4_Week 12 - No change | 6.0 | 5.6 | 14.6 | 4.6
  5_Week 12 - Minimally worse: number analyzed (Participants) | 151 | 144 | 151 | 285
  5_Week 12 - Minimally worse | 2.6 | 4.2 | 0.7 | 1.4
  6_Week 12 - Much worse: number analyzed (Participants) | 151 | 144 | 151 | 285
  6_Week 12 - Much worse | 0.7 | 0.7 | 0.0 | 0.4
  7_Week 12 - Very Much Worse: number analyzed (Participants) | 151 | 144 | 151 | 285
  7_Week 12 - Very Much Worse | 0.7 | 0.0 | 0.0 | 0.7
  1_Week 52 - Very Much Improved: number analyzed (Participants) | 93 | 81 | 105 | 138
  1_Week 52 - Very Much Improved | 34.4 | 35.8 | 24.8 | 37.0
  2_Week 52- Much Improved: number analyzed (Participants) | 93 | 81 | 105 | 138
  2_Week 52- Much Improved | 41.9 | 46.9 | 38.1 | 37.7
  3_Week 52 - Minimally Improved: number analyzed (Participants) | 93 | 81 | 105 | 138
  3_Week 52 - Minimally Improved | 17.2 | 13.6 | 22.9 | 21.7
  4_Week 52 - No change: number analyzed (Participants) | 93 | 81 | 105 | 138
  4_Week 52 - No change | 4.3 | 2.5 | 12.4 | 2.2
  5_Week 52 - Minimally worse: number analyzed (Participants) | 93 | 81 | 105 | 138
  5_Week 52 - Minimally worse | 1.1 | 0.0 | 1.9 | 0.7
  6_Week 52 - Much worse: number analyzed (Participants) | 93 | 81 | 105 | 138
  6_Week 52 - Much worse | 1.1 | 1.2 | 0.0 | 0.0
  7_Week 52 - Very Much Worse: number analyzed (Participants) | 93 | 81 | 105 | 138
  7_Week 52 - Very Much Worse | 0.0 | 0.0 | 0.0 | 0.7

44. Secondary Outcome: Change From Baseline in Mean Endometrial Thickness -- (Efficacy Study Part, Safety Study Part)
Description: Change from baseline for non-hysterectomized subjects by visit (Efficacy Study Part and Safety Study Part).
  Endometrial thickness was assessed by transvaginal ultrasound (TVUS).
Time Frame: Screening, Week 13, 29, 41, 53, Follow-up (Week 55/56), and early discontinuation (up to Week 53 for hysterectomized subjects and Week 55/56 for non-hysterectomized subjects)
Population: Safety Analysis Set (SAF) for Efficacy study part: included all subjects who received at least one dose of randomized study medication. The SAF was used for all safety analyses and background characteristics and all analyses on this set were based on the treatment received.
  Safety Analysis Set (SAF) for Safety study part: included all subjects who received at least one dose of study medication. The SAF was used for all safety analyses and background characteristics.
Measure: Mean (95% Confidence Interval); unit: millimeter
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part | Estetrol 20 mg - Safety Study Part
Number analyzed (Participants) | 93 | 93 | 95 | 229
millimeter
  Week 13: number analyzed (Participants) | 65 | 55 | 68 | 116
  Week 13 | 4.20 [2.66 to 5.74] | 3.90 [2.44 to 5.36] | 0.23 [-0.08 to 0.54] | 6.91 [5.76 to 8.07]
  Week 29: number analyzed (Participants) | 36 | 33 | 57 | 48
  Week 29 | 2.65 [0.88 to 4.43] | 3.62 [1.52 to 5.71] | 0.32 [-0.05 to 0.69] | 4.34 [3.00 to 5.69]
  Week 41: number analyzed (Participants) | 27 | 20 | 38 | 31
  Week 41 | 1.74 [0.77 to 2.72] | 2.08 [0.32 to 3.83] | 0.52 [-0.05 to 1.09] | 3.08 [1.75 to 4.41]
  Week 53: number analyzed (Participants) | 34 | 25 | 42 | 24
  Week 53 | 1.93 [0.40 to 3.45] | 1.66 [0.63 to 2.69] | 0.63 [0.13 to 1.14] | 3.19 [1.70 to 4.68]
  Week 55/56 (Follow-up): number analyzed (Participants) | 59 | 54 | 45 | 134
  Week 55/56 (Follow-up) | 0.84 [0.36 to 1.32] | 1.31 [0.72 to 1.91] | 0.05 [-0.27 to 0.37] | 1.13 [0.76 to 1.51]
  Early Discontinuation: number analyzed (Participants) | 20 | 30 | 11 | 106
  Early Discontinuation | 5.21 [1.26 to 9.16] | 5.56 [3.55 to 7.58] | -0.23 [-1.06 to 0.60] | 4.96 [3.80 to 6.12]

45. Secondary Outcome: Number of Subjects in the Different Endometrial Categories -- (Efficacy Study Part, Safety Study Part)
Description: A summary of the Final/Consensus diagnosis of endometrial biopsies across all post-baseline visits is provided. An endometrial biopsy was obtained during the Screening period and at the EOT/Early Discontinuation visit. An additional unscheduled biopsy could have been taken if a subject presented with endometrial thickness >10 mm on TVUS, or persistent and/or recurrent bleeding.
  Biopsies were read by 3 independent expert pathologists as per regulatory requirements. The Final/Consensus diagnosis was defined as the concurrence of at least 2 diagnoses from the 3 pathologists, and if there was no agreement among at least 2 pathologists, the most severe pathologic diagnosis was used.
  The World Health Organization (WHO) classification which separates endometrial diagnoses into 6 categories (benign endometrium, simple hyperplasia, complex hyperplasia, simple atypical hyperplasia, complex atypical hyperplasia, carcinoma) was applied for the assessment of the Final/Consensus diagnosis.
Time Frame: Screening and Week 53.
Population: Safety Analysis Set (SAF) for Efficacy study part: included all subjects who received at least one dose of randomized study medication. All analyses on this set were based on the treatment received.
  Safety Analysis Set (SAF) for Safety study part: included all subjects who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part | Estetrol 20 mg - Safety Study Part
Number analyzed (Participants) | 93 | 93 | 95 | 229
Participants
  Subjects with performed biopsy | 46 | 48 | 28 | 142
  Subjects with evaluable biopsy: number analyzed (Participants) | 46 | 48 | 28 | 142
  Subjects with evaluable biopsy | 44 | 45 | 20 | 132
  Benign Endometrium: number analyzed (Participants) | 44 | 45 | 20 | 132
  Benign Endometrium | 41 | 40 | 20 | 125
  Simple Hyperplasia Without Atypia: number analyzed (Participants) | 44 | 45 | 20 | 132
  Simple Hyperplasia Without Atypia | 1 | 3 | 0 | 7
  Simple Hyperplasia With Atypia: number analyzed (Participants) | 44 | 45 | 20 | 132
  Simple Hyperplasia With Atypia | 0 | 1 | 0 | 0
  Complex Hyperplasia Without Atypia: number analyzed (Participants) | 44 | 45 | 20 | 132
  Complex Hyperplasia Without Atypia | 1 | 1 | 0 | 0
  Complex Hyperplasia With Atypia: number analyzed (Participants) | 44 | 45 | 20 | 132
  Complex Hyperplasia With Atypia | 1 | 0 | 0 | 0
  Carcinoma: number analyzed (Participants) | 44 | 45 | 20 | 132
  Carcinoma | 0 | 0 | 0 | 0

46. Secondary Outcome: Vaginal Bleeding and/or Spotting During Each 28-day Cycle of Treatment With E4 -- (Efficacy Study Part, Safety Study Part)
Description: Frequency (percentage) of non-hysterectomized participants with vaginal bleeding and/or spotting during each 28-day cycle of treatment with E4, based on the subject diary (Efficacy study part and Safety study part).
  Vaginal bleeding was daily recorded by the participant in the diary. Absence or occurrence of vaginal bleeding/ spotting was assessed using the scale below: 0=Absence of vaginal bleeding or spotting; 1=Spotting: evidence of minimal blood loss requiring none or at most one pad, tampon or panty liner per day; 2=Bleeding: evidence of blood loss requiring more than one pad, tampon or panty liner per day.
Time Frame: Cycle 1,2,3,4,5,6,7,8,9,10,11,12,13
Population: as for outcome 45
Measure: Number; unit: percentage of participants
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part | Estetrol 20 mg - Safety Study Part
Number analyzed (Participants) | 93 | 93 | 95 | 229
percentage of participants
  1_Cycle 1 Subjects with any bleeding and/or spotting during the cycle: number analyzed (Participants) | 85 | 88 | 89 | 203
  1_Cycle 1 Subjects with any bleeding and/or spotting during the cycle | 9.4 | 13.6 | 5.6 | 12.3
  2_Cycle 1 Subjects with spotting only during the cycle: number analyzed (Participants) | 85 | 88 | 89 | 203
  2_Cycle 1 Subjects with spotting only during the cycle | 5.9 | 13.6 | 4.5 | 8.4
  1_Cycle 2 Subjects with any bleeding and/or spotting during the cycle: number analyzed (Participants) | 84 | 83 | 83 | 175
  1_Cycle 2 Subjects with any bleeding and/or spotting during the cycle | 23.8 | 37.3 | 7.2 | 42.3
  2_Cycle 2 Subjects with spotting only during the cycle: number analyzed (Participants) | 84 | 83 | 83 | 175
  2_Cycle 2 Subjects with spotting only during the cycle | 13.1 | 25.3 | 4.8 | 11.4
  1_Cycle 3 Subjects with any bleeding and/or spotting during the cycle: number analyzed (Participants) | 79 | 77 | 77 | 152
  1_Cycle 3 Subjects with any bleeding and/or spotting during the cycle | 36.7 | 50.6 | 1.3 | 59.2
  2_Cycle 3 Subjects with spotting only during the cycle: number analyzed (Participants) | 79 | 77 | 77 | 152
  2_Cycle 3 Subjects with spotting only during the cycle | 10.1 | 19.5 | 0.0 | 19.7
  1_Cycle 4 Subjects with any bleeding and/or spotting during the cycle: number analyzed (Participants) | 71 | 67 | 70 | 117
  1_Cycle 4 Subjects with any bleeding and/or spotting during the cycle | 31.0 | 46.3 | 2.9 | 55.6
  2_Cycle 4 Subjects with spotting only during the cycle: number analyzed (Participants) | 71 | 67 | 70 | 117
  2_Cycle 4 Subjects with spotting only during the cycle | 8.5 | 16.4 | 2.9 | 15.4
  1_Cycle 5 Subjects with any bleeding and/or spotting during the cycle: number analyzed (Participants) | 48 | 47 | 56 | 77
  1_Cycle 5 Subjects with any bleeding and/or spotting during the cycle | 20.8 | 40.4 | 7.1 | 48.1
  2_Cycle 5 Subjects with spotting only during the cycle: number analyzed (Participants) | 48 | 47 | 56 | 77
  2_Cycle 5 Subjects with spotting only during the cycle | 6.3 | 10.6 | 7.1 | 19.5
  1_Cycle 6 Subjects with any bleeding and/or spotting during the cycle: number analyzed (Participants) | 44 | 39 | 55 | 61
  1_Cycle 6 Subjects with any bleeding and/or spotting during the cycle | 15.9 | 46.2 | 1.8 | 36.1
  2_Cycle 6 Subjects with spotting only during the cycle: number analyzed (Participants) | 44 | 39 | 55 | 61
  2_Cycle 6 Subjects with spotting only during the cycle | 4.5 | 20.5 | 0.0 | 19.7
  1_Cycle 7 Subjects with any bleeding and/or spotting during the cycle: number analyzed (Participants) | 42 | 35 | 53 | 53
  1_Cycle 7 Subjects with any bleeding and/or spotting during the cycle | 11.9 | 25.7 | 3.8 | 37.7
  2_Cycle 7 Subjects with spotting only during the cycle: number analyzed (Participants) | 42 | 35 | 53 | 53
  2_Cycle 7 Subjects with spotting only during the cycle | 4.8 | 8.6 | 3.8 | 15.1
  1_Cycle 8 Subjects with any bleeding and/or spotting during the cycle: number analyzed (Participants) | 40 | 33 | 52 | 42
  1_Cycle 8 Subjects with any bleeding and/or spotting during the cycle | 17.5 | 24.2 | 1.9 | 33.3
  2_Cycle 8 Subjects with spotting only during the cycle: number analyzed (Participants) | 40 | 33 | 52 | 42
  2_Cycle 8 Subjects with spotting only during the cycle | 5.0 | 3.0 | 1.9 | 7.1
  1_Cycle 9 Subjects with any bleeding and/or spotting during the cycle: number analyzed (Participants) | 36 | 29 | 50 | 38
  1_Cycle 9 Subjects with any bleeding and/or spotting during the cycle | 13.9 | 17.2 | 0.0 | 31.6
  2_Cycle 9 Subjects with spotting only during the cycle: number analyzed (Participants) | 36 | 29 | 50 | 38
  2_Cycle 9 Subjects with spotting only during the cycle | 2.8 | 6.9 | 0.0 | 15.8
  1_Cycle 10 Subjects with any bleeding and/or spotting during the cycle: number analyzed (Participants) | 35 | 27 | 50 | 30
  1_Cycle 10 Subjects with any bleeding and/or spotting during the cycle | 11.4 | 11.1 | 0.0 | 36.7
  2_Cycle 10 Subjects with spotting only during the cycle: number analyzed (Participants) | 35 | 27 | 50 | 30
  2_Cycle 10 Subjects with spotting only during the cycle | 0.0 | 0.0 | 0.0 | 23.3
  1_Cycle 11 Subjects with any bleeding and/or spotting during the cycle: number analyzed (Participants) | 36 | 26 | 40 | 28
  1_Cycle 11 Subjects with any bleeding and/or spotting during the cycle | 11.1 | 11.5 | 2.5 | 25.0
  2_Cycle 11 Subjects with spotting only during the cycle: number analyzed (Participants) | 36 | 26 | 40 | 28
  2_Cycle 11 Subjects with spotting only during the cycle | 5.6 | 3.8 | 0.0 | 17.9
  1_Cycle 12 Subjects with any bleeding and/or spotting during the cycle: number analyzed (Participants) | 35 | 24 | 40 | 27
  1_Cycle 12 Subjects with any bleeding and/or spotting during the cycle | 5.7 | 16.7 | 2.5 | 29.6
  2_Cycle 12 Subjects with spotting only during the cycle: number analyzed (Participants) | 35 | 24 | 40 | 27
  2_Cycle 12 Subjects with spotting only during the cycle | 2.9 | 12.5 | 2.5 | 18.5
  1_Cycle 13 Subjects with any bleeding and/or spotting during the cycle: number analyzed (Participants) | 31 | 24 | 42 | 21
  1_Cycle 13 Subjects with any bleeding and/or spotting during the cycle | 6.5 | 16.7 | 2.4 | 23.8
  2_Cycle 13 Subjects with spotting only during the cycle: number analyzed (Participants) | 31 | 24 | 42 | 21
  2_Cycle 13 Subjects with spotting only during the cycle | 6.5 | 4.2 | 2.4 | 19.0

47. Secondary Outcome: Number of Days With Bleeding or Spotting by Cycle for Non-Hysterectomized Subjects (Efficacy Study Part, Safety Study Part)
Description: Number of days with bleeding or spotting during each 28-day cycle of treatment for non-hysterectomized (NH) subjects (Efficacy study part, Safety study part). The Overall Number of Participants Analyzed corresponds to the total number of NH participants in each study arm in the SAF. For each cycle, the number analyzed corresponds to the number of NH subjects with corresponding bleeding/spotting information available in the diary for that cycle. Women with bleeding and spotting during a cycle are counted in both the Bleeding Days and Spotting Days categories for that cycle.
  Vaginal bleeding was recorded daily by the participants in the diary. Absence or occurrence of vaginal bleeding/spotting was assessed using the scale below: 0=Absence of vaginal bleeding or spotting; 1=Spotting: evidence of minimal blood loss requiring none or at most one pad, tampon or panty liner per day; 2=Bleeding: evidence of blood loss requiring more than one pad, tampon or panty liner per day.
Time Frame: Cycle 1,2,3,4,5,6,7,8,9,10,11,12,13.
Population: Safety Analysis Set (SAF) for Efficacy study part: included all subjects who received at least one dose of randomized study medication. All analyses on this set based on the treatment received.
  Outcome assessed only in the non-hysterectomized (NH) women of SAF: n=93, 93, 95 in E4 15 mg, E4 20 mg, Placebo, respectively.
  Safety Analysis Set (SAF) for Safety study part: included all subjects who received at least one dose of study medication.
  Outcome assessed only in the NH women of SAF: n=229.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part | Estetrol 20 mg - Safety Study Part
Number analyzed (Participants) | 93 | 93 | 95 | 229
days
  Cycle 1 - No Bleeding, No Spotting: number analyzed (Participants) | 77 | 76 | 84 | 178
  Cycle 1 - No Bleeding, No Spotting | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Cycle 1 - Bleeding Days: number analyzed (Participants) | 3 | 0 | 1 | 8
  Cycle 1 - Bleeding Days | 3.7 (2.08) |  | 4.0 (NA) — Data available from only 1 subject. | 1.0 (0.00)
  Cycle 1 - Spotting Days: number analyzed (Participants) | 7 | 12 | 5 | 23
  Cycle 1 - Spotting Days | 3.3 (2.36) | 1.8 (1.03) | 4.2 (2.68) | 1.0 (0.00)
  Cycle 2 - No Bleeding, No Spotting: number analyzed (Participants) | 64 | 52 | 77 | 101
  Cycle 2 - No Bleeding, No Spotting | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Cycle 2 - Bleeding Days: number analyzed (Participants) | 9 | 10 | 2 | 54
  Cycle 2 - Bleeding Days | 5.3 (4.58) | 4.2 (1.87) | 2.0 (1.41) | 1.1 (0.29)
  Cycle 2 - Spotting Days: number analyzed (Participants) | 20 | 31 | 6 | 70
  Cycle 2 - Spotting Days | 3.8 (3.56) | 4.1 (3.73) | 3.8 (2.14) | 1.1 (0.35)
  Cycle 3 - No Bleeding, No Spotting: number analyzed (Participants) | 50 | 38 | 76 | 62
  Cycle 3 - No Bleeding, No Spotting | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Cycle 3 - Bleeding Days: number analyzed (Participants) | 21 | 24 | 1 | 60
  Cycle 3 - Bleeding Days | 6.0 (4.79) | 8.8 (6.48) | 5.0 (NA) — Data available from only 1 subject. | 1.1 (0.34)
  Cycle 3 - Spotting Days: number analyzed (Participants) | 27 | 38 | 1 | 84
  Cycle 3 - Spotting Days | 6.8 (6.39) | 5.1 (3.49) | 1.0 (NA) — Data available from only 1 subject. | 1.1 (0.31)
  Cycle 4 - No Bleeding, No Spotting: number analyzed (Participants) | 49 | 36 | 68 | 52
  Cycle 4 - No Bleeding, No Spotting | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Cycle 4 - Bleeding Days: number analyzed (Participants) | 16 | 20 | 0 | 47
  Cycle 4 - Bleeding Days | 2.6 (2.19) | 2.7 (2.85) |  | 1.2 (0.38)
  Cycle 4 - Spotting Days: number analyzed (Participants) | 20 | 28 | 2 | 59
  Cycle 4 - Spotting Days | 1.9 (1.59) | 2.1 (1.59) | 1.0 (0.00) | 1.2 (0.47)
  Cycle 5 - No Bleeding, No Spotting: number analyzed (Participants) | 38 | 28 | 52 | 40
  Cycle 5 - No Bleeding, No Spotting | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Cycle 5 - Bleeding Days: number analyzed (Participants) | 7 | 14 | 0 | 22
  Cycle 5 - Bleeding Days | 1.0 (0.00) | 1.0 (0.00) |  | 1.1 (0.35)
  Cycle 5 - Spotting Days: number analyzed (Participants) | 9 | 18 | 4 | 35
  Cycle 5 - Spotting Days | 1.0 (0.00) | 1.0 (0.00) | 1.0 (0.00) | 1.1 (0.36)
  Cycle 6 - No Bleeding, No Spotting: number analyzed (Participants) | 37 | 21 | 54 | 39
  Cycle 6 - No Bleeding, No Spotting | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Cycle 6 - Bleeding Days: number analyzed (Participants) | 5 | 10 | 1 | 10
  Cycle 6 - Bleeding Days | 1.0 (0.00) | 1.1 (0.32) | 1.0 (NA) — Data available from only 1 subject. | 1.1 (0.32)
  Cycle 6 - Spotting Days: number analyzed (Participants) | 6 | 17 | 1 | 19
  Cycle 6 - Spotting Days | 1.0 (0.00) | 1.1 (0.24) | 1.0 (NA) — Data available from only 1 subject. | 1.1 (0.23)
  Cycle 7 - No Bleeding, No Spotting: number analyzed (Participants) | 37 | 26 | 51 | 33
  Cycle 7 - No Bleeding, No Spotting | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Cycle 7 - Bleeding Days: number analyzed (Participants) | 3 | 6 | 0 | 12
  Cycle 7 - Bleeding Days | 1.0 (0.00) | 1.2 (0.41) |  | 1.2 (0.39)
  Cycle 7 - Spotting Days: number analyzed (Participants) | 4 | 9 | 2 | 18
  Cycle 7 - Spotting Days | 1.0 (0.00) | 1.1 (0.33) | 1.0 (0.00) | 1.2 (0.38)
  Cycle 8 - No Bleeding, No Spotting: number analyzed (Participants) | 33 | 25 | 51 | 28
  Cycle 8 - No Bleeding, No Spotting | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Cycle 8 - Bleeding Days: number analyzed (Participants) | 5 | 7 | 0 | 11
  Cycle 8 - Bleeding Days | 1.2 (0.45) | 1.3 (0.49) |  | 1.1 (0.30)
  Cycle 8 - Spotting Days: number analyzed (Participants) | 6 | 7 | 1 | 13
  Cycle 8 - Spotting Days | 1.2 (0.41) | 1.4 (0.53) | 1.0 (NA) — Data available from only 1 subject. | 1.1 (0.28)
  Cycle 9 - No Bleeding, No Spotting: number analyzed (Participants) | 31 | 24 | 50 | 26
  Cycle 9 - No Bleeding, No Spotting | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Cycle 9 - Bleeding Days: number analyzed (Participants) | 4 | 3 | 0 | 6
  Cycle 9 - Bleeding Days | 1.0 (0.00) | 1.0 (0.00) |  | 1.2 (0.41)
  Cycle 9 - Spotting Days: number analyzed (Participants) | 4 | 3 | 0 | 12
  Cycle 9 - Spotting Days | 1.0 (0.00) | 1.0 (0.00) |  | 1.0 (0.00)
  Cycle 10 - No Bleeding, No Spotting: number analyzed (Participants) | 31 | 24 | 50 | 19
  Cycle 10 - No Bleeding, No Spotting | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Cycle 10 - Bleeding Days: number analyzed (Participants) | 4 | 3 | 0 | 4
  Cycle 10 - Bleeding Days | 1.0 (0.00) | 1.0 (0.00) |  | 1.3 (0.50)
  Cycle 10 - Spotting Days: number analyzed (Participants) | 4 | 2 | 0 | 11
  Cycle 10 - Spotting Days | 1.0 (0.00) | 1.0 (0.00) |  | 1.0 (0.00)
  Cycle 11 - No Bleeding, No Spotting: number analyzed (Participants) | 32 | 23 | 39 | 21
  Cycle 11 - No Bleeding, No Spotting | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Cycle 11 - Bleeding Days: number analyzed (Participants) | 2 | 2 | 1 | 2
  Cycle 11 - Bleeding Days | 1.0 (0.00) | 1.0 (0.00) | 1.0 | 1.5 (0.71)
  Cycle 11 - Spotting Days: number analyzed (Participants) | 4 | 2 | 1 | 7
  Cycle 11 - Spotting Days | 1.0 (0.00) | 1.0 (0.00) | 1.0 (NA) — Data available from only 1 subject. | 1.1 (0.38)
  Cycle 12 - No Bleeding, No Spotting: number analyzed (Participants) | 33 | 20 | 39 | 19
  Cycle 12 - No Bleeding, No Spotting | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Cycle 12 - Bleeding Days: number analyzed (Participants) | 1 | 1 | 0 | 3
  Cycle 12 - Bleeding Days | 1.0 (NA) — Data available from only 1 subject. | 1.0 (NA) — Data available from only 1 subject. |  | 1.3 (0.58)
  Cycle 12 - Spotting Days: number analyzed (Participants) | 2 | 4 | 1 | 8
  Cycle 12 - Spotting Days | 1.0 (0.00) | 1.0 (0.00) | 1.0 (NA) — Data available from only 1 subject. | 1.1 (0.35)
  Cycle 13 - No Bleeding, No Spotting: number analyzed (Participants) | 29 | 20 | 41 | 16
  Cycle 13 - No Bleeding, No Spotting | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Cycle 13 - Bleeding Days: number analyzed (Participants) | 0 | 3 | 0 | 1
  Cycle 13 - Bleeding Days |  | 1.0 (0.00) |  | 1.0 (NA) — Data available from only 1 subject.
  Cycle 13 - Spotting Days: number analyzed (Participants) | 2 | 4 | 1 | 5
  Cycle 13 - Spotting Days | 1.0 (0.00) | 1.0 (0.00) | 1.0 (NA) — Data available from only 1 subject. | 1.2 (0.45)

48. Secondary Outcome: Cumulative Rate of Amenorrhea (Absence of Any Bleeding or Spotting) During Each 28-day Cycle of Treatment With E4 -- (Efficacy Study Part, Safety Study Part)
Description: Cumulative rates of amenorrhea defined as the percentage of women who reported consecutive cycles of amenorrhea (absence of any bleeding or spotting) for a given cycle of time (Efficacy study part and Safety study part).
  Percentages (%) are based on the number of non-hysterectomized subjects with amenorrhea diary data available through cycle 13 in the Safety Analysis Set in each treatment arm.
Time Frame: Cycle 1,2,3,4,5,6,7,8,9,10,11,12,13.
Population: as for outcome 45
Measure: Number; unit: percentage of participants
Arm/Group | Estetrol 15 mg - Efficacy Study Part | Estetrol 20 mg - Efficacy Study Part | Placebo - Efficacy Study Part | Estetrol 20 mg - Safety Study Part
Number analyzed (Participants) | 82 | 83 | 88 | 229
percentage of participants
  Cycle 1-13 | 34.4 | 25.8 | 66.3 | 18.8
  Cycle 2-13 | 35.5 | 28.0 | 66.3 | 20.5
  Cycle 3-13 | 37.6 | 31.2 | 69.5 | 25.3
  Cycle 4-13 | 40.9 | 36.6 | 69.5 | 30.6
  Cycle 5-13 | 44.1 | 37.6 | 70.5 | 32.3
  Cycle 6-13 | 45.2 | 37.6 | 71.6 | 33.6
  Cycle 7-13 | 46.2 | 41.9 | 71.6 | 33.6
  Cycle 8-13 | 46.2 | 44.1 | 74.7 | 34.9
  Cycle 9-13 | 46.2 | 45.2 | 77.9 | 35.4
  Cycle 10-13 | 49.5 | 46.2 | 77.9 | 35.8
  Cycle 11-13 | 52.7 | 46.2 | 77.9 | 36.7
  Cycle 12-13 | 53.8 | 46.2 | 81.1 | 36.7
  Cycle 13 | 53.8 | 46.2 | 83.2 | 37.1

49. Secondary Outcome: Number of Participants With Serious Adverse Events (SAE) in SOC 'Reproductive System and Breast Disorders' or With PT 'Abdominal Pain' by Hysterectomy Status (Hysterectomized and Non-Hysterectomized) -- (Efficacy Study Part, Safety Study Part)
Description: Number of participants with SAEs belonging to the system organ class (SOC) 'Reproductive system and breast disorders' or with preferred term (PT) 'Abdominal Pain', by hysterectomy status (hysterectomized and non-hysterectomized); Efficacy Study Part and Safety Study Part.
  Adverse events (AEs) are defined as occurring from time of first IMP intake until last visit or any event already present that worsens (in either intensity or frequency) after exposure to the treatment.
  AEs in SOC 'Reproductive System and Breast Disorders' or with PT 'Abdominal Pain' were reported separately for non-hysterectomized (NH) and hysterectomized women. For endometrial protection, NH women received commercially available P4 200 mg once daily for 14 consecutive days, after completing the E4/placebo treatment. All AEs were collected until the last visit, including the period of P4 intake, and reported grouped by arm (ESP: E4 15 mg/E4 20 mg/Placebo; SSP: E4 20 mg).
Time Frame: Day 1 (allocation to treatment) until Week 53 (hysterectomized participants) or Week 55/56 (non-hysterectomized participants).
Population: Safety Analysis Set (SAF) for Efficacy study part: included all randomized subjects who received at least one dose of randomized study medication. All analyses on this set were based on the treatment received.
  Safety Analysis Set (SAF) for Safety study part: included all subjects who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- Estetrol 15 mg -- Hysterectomized -- Efficacy Study Part; Estetrol 15 mg -- Non-Hysterectomized -- Efficacy Study Part: Estetrol (E4) 15 mg oral tablet, administered once daily for up to 53 weeks.
- Estetrol 20 mg -- Hysterectomized -- Efficacy Study Part; Estetrol 20 mg -- Non-Hysterectomized -- Efficacy Study Part; Estetrol 20 mg -- Hysterectomized -- Safety Study Part; Estetrol 20 mg -- Non-Hysterectomized -- Safety Study Part: Estetrol (E4) 20 mg oral tablet, administered once daily for up to 53 weeks.
- Placebo -- Hysterectomized -- Efficacy Study Part; Placebo -- Non-Hysterectomized -- Efficacy Study Part: Placebo was administered orally once daily for up to 53 weeks.
Arm/Group | Estetrol 15 mg -- Hysterectomized -- Efficacy Study Part | Estetrol 15 mg -- Non-Hysterectomized -- Efficacy Study Part | Estetrol 20 mg -- Hysterectomized -- Efficacy Study Part | Estetrol 20 mg -- Non-Hysterectomized -- Efficacy Study Part | Placebo -- Hysterectomized -- Efficacy Study Part | Placebo -- Non-Hysterectomized -- Efficacy Study Part | Estetrol 20 mg -- Hysterectomized -- Safety Study Part | Estetrol 20 mg -- Non-Hysterectomized -- Safety Study Part
Number analyzed (Participants) | 99 | 93 | 100 | 93 | 99 | 95 | 201 | 229
Participants
  Reproductive System and Breast Disorders | 0 | 15 | 0 | 20 | 0 | 0 | 1 | 53
  Ovarian vein thrombosis | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Endometrial disorder | 0 | 12 | 0 | 12 | 0 | 0 | 0 | 45
  Endometrial hyperplasia | 0 | 3 | 0 | 8 | 0 | 0 | 0 | 6
  Vaginal haemorrhage | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3

50. Secondary Outcome: Number of Participants With Non-serious Adverse Events (AEs) in SOC 'Reproductive System and Breast Disorders' or With PT 'Abdominal Pain' by Hysterectomy Status -- (Efficacy Study Part, Safety Study Part)
Description: Number of participants with non-serious AEs at 2% threshold in any treatment group in the system organ class (SOC) 'Reproductive system and breast disorders' or with preferred term (PT) 'Abdominal Pain', during the Efficacy Study Part and the Safety Study Part.
  Adverse events (AEs) are defined as occurring from time of first IMP intake until last visit or any event already present that worsens (in either intensity or frequency) after exposure to the treatment.
  AEs in SOC 'Reproductive System and Breast Disorders' or with PT 'Abdominal Pain' were reported separately for non-hysterectomized (NH) and hysterectomized women. For endometrial protection, NH women received commercially available P4 200 mg once daily for 14 consecutive days, after completing the E4/placebo treatment. All AEs were collected until the last visit, including the period of P4 intake, and reported grouped by arm (ESP: E4 15 mg/E4 20 mg/Placebo; SSP: E4 20 mg).
Time Frame: as for outcome 49
Population: as for outcome 49
Measure: Count of Participants; unit: Participants
Arm/Group | Estetrol 15 mg -- Non-Hysterectomized -- Efficacy Study Part | Estetrol 15 mg -- Hysterectomized -- Efficacy Study Part | Estetrol 20 mg -- Non-Hysterectomized -- Efficacy Study Part | Estetrol 20 mg -- Hysterectomized -- Efficacy Study Part | Placebo -- Non-Hysterectomized -- Efficacy Study Part | Placebo -- Hysterectomized -- Efficacy Study Part | Estetrol 20 mg -- Non-Hysterectomized -- Safety Study Part | Estetrol 20 mg -- Hysterectomized -- Safety Study Part
Number analyzed (Participants) | 93 | 99 | 93 | 100 | 95 | 99 | 229 | 201
Participants
  Reproductive system and breast disorders | 43 | 25 | 52 | 22 | 12 | 9 | 166 | 57
  Vaginal haemorrhage | 28 | 0 | 35 | 0 | 5 | 0 | 103 | 1
  Endometrial thickening | 15 | 0 | 18 | 0 | 1 | 0 | 59 | 0
  Endometrial disorder | 9 | 0 | 11 | 0 | 1 | 0 | 40 | 0
  Breast tenderness | 7 | 15 | 10 | 14 | 0 | 6 | 34 | 28
  Vaginal discharge | 7 | 2 | 1 | 2 | 1 | 0 | 14 | 5
  Uterine haemorrhage | 4 | 0 | 4 | 0 | 0 | 0 | 11 | 0
  Uterine spasm | 2 | 0 | 4 | 0 | 0 | 1 | 15 | 0
  Ovarian cyst | 0 | 1 | 2 | 1 | 3 | 1 | 0 | 2
  Endometrial hyperplasia | 1 | 0 | 3 | 0 | 0 | 0 | 4 | 0
  Nipple pain | 2 | 3 | 2 | 4 | 0 | 2 | 14 | 14
  Menopausal symptoms | 2 | 1 | 1 | 0 | 0 | 1 | 4 | 3
  Vulvovaginal discomfort | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Breast pain | 0 | 2 | 1 | 2 | 0 | 1 | 2 | 7
  Breast discomfort | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 5
  Gastrointestinal disorders / PT Abdominal pain lower | 0 | 1 | 0 | 3 | 0 | 1 | 4 | 0
  Gastrointestinal disorders / PT Abdominal pain | 2 | 2 | 3 | 2 | 2 | 0 | 17 | 3
  Gastrointestinal disorders / PT Abdominal pain upper | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 (allocation to treatment) until Week 53 (hysterectomized participants) or Week 55/56 (non-hysterectomized participants)
Description: AEs were reported by arm (ESP:E4 15 mg;E4 20 mg;placebo, and SSP:E4 20 mg); AEs in the SOC Reproductive System and Breast Disorders or PT Abdominal Pain were analyzed by hysterectomy status (see Secondary Outcomes 49-50). NH participants took P4 200 mg for 14 days after completion of E4/placebo treatment, for endometrial protection. AEs collected during P4 treatment were included in the E4 or placebo arm to which the participant was allocated; a separate analysis of these AEs was not performed.
Groups:
- Estetrol 15 mg - Efficacy Part: Estetrol (E4) 15 mg oral tablet, administered once daily for up to 53 weeks.
- Estetrol 20 mg - Efficacy Part; Estetrol 20 mg - Safety Part: Estetrol (E4) 20 mg oral tablet, administered once daily for up to 53 weeks.
- Placebo - Efficacy Part: Placebo was administered orally once daily for up to 53 weeks.
Arm/Group | Estetrol 15 mg - Efficacy Part | Estetrol 20 mg - Efficacy Part | Placebo - Efficacy Part | Estetrol 20 mg - Safety Part
All-Cause Mortality (participants affected / at risk) | 1/192 | 0/193 | 0/194 | 0/430
Serious Adverse Events (participants affected / at risk) | 21/192 | 21/193 | 3/194 | 60/430
Other Adverse Events (participants affected / at risk) | 125/192 | 126/193 | 98/194 | 309/430
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estetrol 15 mg - Efficacy Part (N=192) | Estetrol 20 mg - Efficacy Part (N=193) | Placebo - Efficacy Part (N=194) | Estetrol 20 mg - Safety Part (N=430)
Endometrial disorder (Reproductive system and breast disorders) | 12 (12) | 12 (12) | 0 (0) | 45 (46)
Endometrial hyperplasia (Reproductive system and breast disorders) | 3 (3) | 8 (8) | 0 (0) | 6 (6)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Ovarian vein thrombosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estetrol 15 mg - Efficacy Part (N=192) | Estetrol 20 mg - Efficacy Part (N=193) | Placebo - Efficacy Part (N=194) | Estetrol 20 mg - Safety Part (N=430)
Vaginal haemorrhage (Reproductive system and breast disorders) | 28 (47) | 35 (56) | 5 (7) | 104 (175)
Breast tenderness (Reproductive system and breast disorders) | 22 (23) | 24 (24) | 6 (6) | 62 (62)
Endometrial thickening (Reproductive system and breast disorders) | 15 (16) | 18 (19) | 1 (1) | 59 (59)
Endometrial disorder (Reproductive system and breast disorders) | 9 (9) | 11 (11) | 1 (1) | 40 (40)
Nipple pain (Reproductive system and breast disorders) | 5 (5) | 6 (6) | 2 (3) | 28 (29)
Vaginal discharge (Reproductive system and breast disorders) | 9 (9) | 3 (3) | 1 (1) | 19 (19)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 4 (4) | 5 (5)
Uterine haemorrhage (Reproductive system and breast disorders) | 4 (4) | 4 (4) | 0 (0) | 11 (12)
Uterine spasm (Reproductive system and breast disorders) | 2 (2) | 4 (4) | 1 (1) | 15 (17)
Breast pain (Reproductive system and breast disorders) | 2 (2) | 3 (3) | 1 (1) | 9 (10)
COVID-19 (Infections and infestations) | 3 (3) | 6 (6) | 5 (5) | 15 (15)
Urinary tract infection (Infections and infestations) | 4 (6) | 5 (5) | 3 (3) | 6 (7)
Sinusitis (Infections and infestations) | 5 (5) | 2 (2) | 3 (3) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 4 (4) | 4 (4) | 8 (8)
Nausea (Gastrointestinal disorders) | 7 (8) | 4 (4) | 2 (2) | 15 (15)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 5 (5) | 2 (2) | 20 (20)
Constipation (Gastrointestinal disorders) | 4 (4) | 4 (5) | 3 (3) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 2 (2) | 3 (3) | 8 (9)
Headache (Nervous system disorders) | 9 (10) | 10 (11) | 19 (21) | 22 (26)
Dizziness (Nervous system disorders) | 5 (5) | 1 (1) | 2 (2) | 9 (10)
Anxiety (Psychiatric disorders) | 6 (6) | 8 (8) | 9 (9) | 5 (6)
Insomnia (Psychiatric disorders) | 5 (5) | 2 (2) | 1 (1) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 7 (7) | 9 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 3 (3) | 3 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (3) | 9 (9)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (4) | 7 (7) | 4 (5)
Weight increased (Investigations) | 5 (5) | 2 (2) | 6 (6) | 16 (16)
Vitamin D deficiency (Metabolism and nutrition disorders) | 5 (5) | 6 (6) | 5 (5) | 0 (0)
Fatigue (General disorders) | 0 (0) | 4 (5) | 6 (6) | 10 (10)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Study Protocol (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT04090957/Prot_000.pdf
  • Statistical Analysis Plan: Efficacy Study Part (ESP) (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT04090957/SAP_001.pdf
  • Statistical Analysis Plan: Safety Study Part (SSP) (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT04090957/SAP_002.pdf